CLINICAL TRIAL: NCT02055118
Title: A Controlled, Randomized, Two-arm, Open-label, Assessor-blinded, Multicenter Study of Intrathecal Idursulfase-IT Administered in Conjunction With Elaprase® in Pediatric Patients With Hunter Syndrome and Early Cognitive Impairment
Brief Title: Study of Intrathecal Idursulfase-IT Administered in Conjunction With Elaprase® in Pediatric Patients With Hunter Syndrome and Early Cognitive Impairment
Acronym: AIM-IT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-HIT-094; 2013-002885-38 (EudraCT Number)
Record Dates: First submitted 2014-01-17; First posted 2014-02-04 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Hunter Syndrome
Keywords: hunters disease; MPS II; lysosomal storage disorder; hunters syndrome; ert treatment; hunter's disease; iduronate sulfatase; MPS society; mps 2; enlarged adenoids; hunter's syndrome; iduronate 2 sulfatase; chronic ear infection; mucopolysaccharides; hunter syndrome therapy; hunter's syndrome treatment; enzyme replacement therapy; hunter syndrome treatment; elaprase; MPSII; lysosomal storage disease; mps diagnosis; mps symptoms; idursulfase; hunter disease; hunter's disease treatment; MPS2
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- idursulfase-IT (Experimental): 10 mg administered via IT using IDDD (intrathecal drug delivery device) once a month for 52 weeks.
  Interventions: Biological: idursulfase-IT
- Nontreatment control (Other): Patients will receive weekly standard of care treatment with IV Elaprase only.
  Interventions: Other: No IT treatment

INTERVENTIONS:
Biological: idursulfase-IT — 10mg
  Arms: idursulfase-IT
Other: No IT treatment — Standard of Care
  Other Names: Non-treatment Control
  Arms: Nontreatment control

SUMMARY:
Study HGT-HIT-094 is a multicenter study designed to determine the effect on clinical parameters of neurodevelopmental status of monthly IT administration of idursulfase-IT 10 mg for 12 months in pediatric patients with Hunter syndrome and cognitive impairment who have previously received and tolerated a minimum of 4 months of therapy with Elaprase.

DETAILED DESCRIPTION:
Elaprase, a large molecular protein, is not expected to cross the blood brain barrier when administered intravenously. A revised formulation of idursulfase, idursulfase-IT, that differs from that of the intravenous (IV) formulation, Elaprase, has been developed to be suitable for delivery into the cerebrospinal fluid (CSF) via intrathecal administration.

Mucopolysaccharidosis II (MPS II) is a rare, X-linked, inherited disease that affects males nearly exclusively. The disease is caused by the absence of, or deficiency in, the activity of the lysosomal enzyme, iduronate-2-sulfatase (I2S) which acts to cleave O-linked sulfate moieties from the glycosaminoglycan (GAG) molecules dermatan sulfate and heparan sulfate.

Study HGT-HIT-094 is a controlled, randomized, two-arm, open-label, assessor-blinded, multicenter study to determine the effect on clinical parameters of neurodevelopmental status of monthly IT administration of idursulfase-IT 10 mg for 12 months in pediatric patients with Hunter syndrome and cognitive impairment who have previously received and tolerated a minimum of 4 months of therapy with Elaprase.

Pediatric patients under 3 years of age will be enrolled into a separate substudy to evaluate the safety and efficacy of idursulfase-IT. The separate substudy is open label and single arm. Patients who are enrolled in the substudy will receive idursulfase-IT treatment and follow the same schedule of study visits.

ELIGIBILITY:
Inclusion Criteria Inclusion Criteria for the Pivotal Study

Patients must meet all of the following criteria to be considered eligible for randomization in the pivotal study:

1. The patient is male and is ≥3 and <18 years of age at the time of informed consent.

   (Patients who are younger than 3 years of age may be enrolled in a separate substudy provided that they meet other inclusion criteria, provided below.)
2. The patient must have a documented diagnosis of MPS II.
3. The patient has evidence at Screening of Hunter syndrome-related cognitive impairment defined as follows:

   A patient who is ≥3 and <13 years of age must have one of the following criteria (3a OR 3b):
   1. A GCA score ≥55 and ≤85 OR
   2. If the patient has a GCA score at Screening >85, there must be evidence of a decrease in GCA score of ≥10 points over 12 months from a previously documented test result in observational study HGT-HIT-090.

      A patient who is ≥13 and <18 years of age must have both of the following criteria (3c AND 3d):
   3. A GCA score of ≥55 and ≤85. AND
   4. There must be evidence of a decrease in GCA score of ≥10 points over 12 months from a previously documented
4. The patient has received and tolerated a minimum of 4 months of therapy with Elaprase during the period immediately prior to Screening.
5. The patient must have sufficient auditory capacity, with a hearing aid(s), if needed, in the Investigator's judgment to complete the required protocol testing and must be compliant with wearing the hearing aid(s), if needed, on scheduled testing days.
6. The patient's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the patient's parent(s) or legally authorized guardian(s) and the patient's assent, if applicable, must be obtained prior to the start of any study procedures.

Inclusion Criteria for the Substudy

Patients must meet all of the following criteria to be considered eligible for enrollment in the separate substudy:

1. The patient is male and is <3 years of age at the time of informed consent.
2. The patient must have a documented diagnosis of MPS II.
3. The patient has evidence at Screening of Hunter syndrome-related cognitive impairment
4. The patient has received and tolerated a minimum of 4 months of therapy with Elaprase during the period immediately prior to Screening.
5. The patient must have sufficient auditory capacity, with a hearing aid(s), if needed, in the Investigator's judgment to complete the required protocol testing and must be compliant with wearing the hearing aid(s), if needed, on scheduled testing days.
6. The patient's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board/Independent Ethics Committee approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the patient's parent(s) or legally authorized guardian(s) must be obtained prior to the start of any study procedures.

Exclusion Criteria

Patients who meet any of the following criteria are not eligible to be randomized into the pivotal study or enrolled in the separate substudy:

1. The patient has clinically significant non-Hunter syndrome-related CNS involvement (such as Fragile-X syndrome) which is judged by the Investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments.
2. The patient has a large chromosomal deletion or complex rearrangement that includes a deletion of the FMR1 and/or FMR2 genes.
3. The patient has a significant medical or psychiatric comorbidity(ies) that might affect study data or confound the integrity of study results.
4. The patient has contra-indications for performance of lumbar puncture such as musculoskeletal/spinal abnormalities or risk of abnormal bleeding.
5. The patient has a history of complications from previous lumbar punctures or technical challenges in conducting lumbar punctures such that the potential risks would exceed possible benefits for the patient.
6. The patient has an opening CSF pressure upon lumbar puncture that exceeds 30.0 cm H2O.
7. The patient has experienced infusion-related anaphylactoid event(s) or has evidence of consistent severe adverse events related to treatment with Elaprase which, in the Investigator's opinion, may pose an unnecessary risk to the patient.
8. The patient has received a cord blood or bone marrow transplant at any time or has received blood product transfusions within 90 days prior to Screening.
9. The patient has a history of poorly controlled seizure disorder.
10. The patient is unable to comply with the protocol (eg, has significant hearing or vision impairment, a clinically relevant medical condition making implementation of the protocol difficult, unstable social situation, known clinically significant psychiatric/behavioral instability, is unable to return for safety evaluations, or is otherwise unlikely to complete the study), as determined by the Investigator.
11. The patient is enrolled in another clinical study that involves clinical investigation or use of any investigational product (drug or [intrathecal/spinal] device) within 30 days prior to study enrollment or at any time during the study.
12. The patient has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to compromised airways or other conditions.
13. The patient has a condition that is contraindicated as described in the SOPH-A-PORT Mini S IDDD Instructions for Use (IFU), including but not limited to the presence of a CSF shunt device in the patient.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (3):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
- Women's and Children's Hospital, 72 King William Road, North Adelaide, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Hôpital Femme Mère Enfant, Bron, France
- Instituto Nacional de Pediatría, Coyoacán, Mexico City, Mexico
- Hospital Infantil Universitario Niño Jesus, Madrid, Spain
- Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Yee KS, Chirila C, Davenport E, Mladsi D, Barnett C, Kronenberger WG. A post hoc analysis of Projected Retained Ability Scores (PRAS) for the longitudinal assessment of cognitive functioning in patients with neuronopathic mucopolysaccharidosis II receiving intrathecal idursulfase-IT. Orphanet J Rare Dis. 2023 Nov 2;18(1):343. doi: 10.1186/s13023-023-02957-2. PMID 37915038
- [Derived] Muenzer J, Burton BK, Harmatz P, Gutierrez-Solana LG, Ruiz-Garcia M, Jones SA, Guffon N, Inbar-Feigenberg M, Bratkovic D, Hale M, Wu Y, Yee KS, Whiteman DAH, Alexanderian D; HGT-HIT-094 Study Group. Intrathecal idursulfase-IT in patients with neuronopathic mucopolysaccharidosis II: Results from a phase 2/3 randomized study. Mol Genet Metab. 2022 Sep-Oct;137(1-2):127-139. doi: 10.1016/j.ymgme.2022.07.017. Epub 2022 Aug 2. PMID 36027721
- [Derived] Muenzer J, Burton BK, Harmatz P, Gutierrez-Solana LG, Ruiz-Garcia M, Jones SA, Guffon N, Inbar-Feigenberg M, Bratkovic D, Hale M, Wu Y, Yee KS, Whiteman DAH, Alexanderian D; SHP609-302 study group. Long-term open-label extension study of the safety and efficacy of intrathecal idursulfase-IT in patients with neuronopathic mucopolysaccharidosis II. Mol Genet Metab. 2022 Sep-Oct;137(1-2):92-103. doi: 10.1016/j.ymgme.2022.07.016. Epub 2022 Aug 2. PMID 35961250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 9 centers in Australia, Canada, France, Mexico, Spain, the United Kingdom and the United States between 24 Mar 2014 (first participant first visit) and 28 Sep 2017 (last participant last visit).
Pre-assignment Details: Overall, 103 participants were screened, of them 54 participants failed to meet the randomization and remaining 49 participants were randomized to receive either IT treatment or No IT treatment in pivotal study. A total of 9 participants were enrolled into the substudy.
Groups:
- No IT Treatment: Participants aged 3 to less than (<) 18 years received Elaprase therapy as standard of care for 12 months.
- IT Treatment: Participants aged 3 to < 18 years received intrathecal (IT) injections of 10 milligram (mg) Idursulfase-IT once monthly for 12 months through SOPH-A-PORT Mini S intrathecal drug delivery device (IDDD) along with Elaprase.
- Substudy: Participants aged less than 3 years received Idursulfase-IT monthly once for 12 months along with Elaprase at a dose of 5 mg if aged less than or equal to (<=) 8 months; 7.5 mg if aged greater than (>) 8 to 30 months and 10 mg if aged > 30 months to 3 years.
Period: Overall Study
Arm/Group | No IT Treatment | IT Treatment | Substudy
Started | 15 | 34 | 9
Completed | 15 | 32 | 9
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants.
Groups:
- No IT Treatment: Participants aged 3 to < 18 years received Elaprase therapy as standard of care for 12 months.
- IT Treatment: Participants aged 3 to < 18 years received IT injections of 10 mg Idursulfase-IT once monthly for 12 months through SOPH-A-PORT Mini S IDDD along with Elaprase.
- Substudy: Participants aged less than 3 years received Idursulfase-IT monthly once for 12 months along with Elaprase at a dose of 5 mg if aged <= 8 months; 7.5 mg if aged > 8 to 30 months and 10 mg if aged > 30 months to 3 years.
- Total: Total of all reporting groups
Arm/Group | No IT Treatment | IT Treatment | Substudy | Total
Number analyzed (Participants) | 15 | 34 | 9 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.29 (2.624) | 4.95 (1.496) | 2.48 (0.483) | 4.65 (1.980)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 15 | 34 | 9 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 1 | 15
  Not Hispanic or Latino | 8 | 25 | 8 | 41
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 4 | 0 | 4
  Race: Black or African American | 0 | 1 | 1 | 2
  Race: White | 12 | 23 | 7 | 42
  Race: Other | 3 | 6 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Differential Ability Scales, Second Edition (DAS-II) General Conceptual Ability (GCA) Standard Score at Week 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The GCA standard score of the DAS-II was used to obtain a general measure of cognitive ability. The GCA score represent a score (mean = 100 and standard deviation of 15) on which higher scores indicate a higher level of cognitive ability. The score ranges from 30 to 170. A positive change value indicates improvement in cognitive ability.
Time Frame: Baseline, Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 29
Score on a scale | -7.4 (4.22) | -4.4 (3.14)
Statistical Analysis 1: Comparison: No IT Treatment vs IT Treatment; The Mixed model repeated measures included fixed categorical effects for treatment, visit week, treatment by visit week interaction, baseline GCA classification factor (less than or equal to [<=] 70 or >70), baseline age group (<6 years or >=6 years), treatment by baseline GCA classification factor interaction, treatment by baseline age group interaction, interaction between baseline GCA classification factor and baseline age group, genotype, and the baseline GCA score as a continuous covariate; Test type: Superiority; p = 0.5669, Mixed model repeated measures; Least squares mean = 3.0, 95% CI 2-sided [-7.3 to 13.3], Standard Error of Mean 5.12

2. Secondary Outcome: Change From Baseline in the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) Adaptive Behavior Composite (ABC) Score at Week 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The ABC score ranges from 20 to 160 on which higher scores indicate a higher level of adaptive functioning. A positive change value indicates improvement in adaptive functioning.
Time Frame: Baseline, Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 14 | 31
Score on a scale | -5.3 (2.55) | -5.0 (2.05)

3. Secondary Outcome: Change From Baseline in the Differential Ability Scales, Second Edition (DAS-II) General Conceptual Ability (GCA) Standard Score at Weeks 16, 28 and 40
Description: as for outcome 1
Time Frame: Baseline, Week 16, Week 28 and Week 40
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: number analyzed (Participants) | 14 | 30
  Week 16 | -2.9 (3.33) | -0.6 (2.54)
  Week 28: number analyzed (Participants) | 12 | 30
  Week 28 | -6.1 (3.34) | -0.3 (2.56)
  Week 40: number analyzed (Participants) | 15 | 30
  Week 40 | -6.4 (3.87) | -3.2 (2.92)

4. Secondary Outcome: Change From Baseline in the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) Adaptive Behavior Composite (ABC) Score at Week 16, 28 and 40
Description: as for outcome 2
Time Frame: Baseline, Week 16, Week 28 and Week 40
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: number analyzed (Participants) | 15 | 31
  Week 16 | -2.8 (2.21) | -3.1 (1.86)
  Week 28: number analyzed (Participants) | 15 | 29
  Week 28 | -1.1 (2.45) | -1.8 (2.01)
  Week 40: number analyzed (Participants) | 14 | 30
  Week 40 | -3.3 (2.41) | -4.7 (1.97)

5. Secondary Outcome: Change From Baseline in Differential Ability Scales, Second Edition (DAS-II) Cluster Standard Scores at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The cluster scores represent a score (mean = 100 and standard deviation of 15) on which higher scores indicate a higher level of cognitive ability in each cluster: verbal (score range: 31-169), nonverbal (score range: 31-166) and spatial (score range: 32-170).
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: Verbal: number analyzed (Participants) | 15 | 32
  Week 16: Verbal | -1.1 (3.75) | -6.9 (2.81)
  Week 16: Nonverbal: number analyzed (Participants) | 14 | 32
  Week 16: Nonverbal | -6.7 (5.06) | 2.6 (3.82)
  Week 16: Spatial: number analyzed (Participants) | 11 | 28
  Week 16: Spatial | -5.6 (3.18) | 1.9 (2.47)
  Week 16: Special Nonverbal Composite (SNC): number analyzed (Participants) | 11 | 28
  Week 16: Special Nonverbal Composite (SNC) | -7.4 (3.95) | -0.7 (2.96)
  Week 28: Verbal: number analyzed (Participants) | 12 | 30
  Week 28: Verbal | -7.0 (4.26) | -5.1 (3.10)
  Week 28: Nonverbal: number analyzed (Participants) | 12 | 30
  Week 28: Nonverbal | -8.8 (5.41) | 0.7 (4.06)
  Week 28: Spatial: number analyzed (Participants) | 9 | 27
  Week 28: Spatial | -7.8 (3.66) | -0.8 (2.70)
  Week 28: Special Nonverbal Composite (SNC): number analyzed (Participants) | 9 | 27
  Week 28: Special Nonverbal Composite (SNC) | -8.0 (4.01) | -1.7 (3.00)
  Week 40: Verbal: number analyzed (Participants) | 15 | 30
  Week 40: Verbal | -7.3 (4.01) | -10.8 (3.07)
  Week 40: Nonverbal: number analyzed (Participants) | 15 | 30
  Week 40: Nonverbal | -8.7 (5.35) | -2.8 (4.09)
  Week 40: Spatial: number analyzed (Participants) | 11 | 27
  Week 40: Spatial | -7.3 (4.39) | 0.6 (3.13)
  Week 40: Special Nonverbal Composite (SNC): number analyzed (Participants) | 11 | 27
  Week 40: Special Nonverbal Composite (SNC) | -9.7 (5.51) | -3.1 (3.78)
  Week 52: Verbal: number analyzed (Participants) | 15 | 30
  Week 52: Verbal | -5.7 (4.45) | -9.8 (3.31)
  Week 52: Nonverbal: number analyzed (Participants) | 15 | 30
  Week 52: Nonverbal | -11.2 (5.61) | -1.5 (4.25)
  Week 52: Spatial: number analyzed (Participants) | 11 | 26
  Week 52: Spatial | -9.6 (4.21) | -4.8 (3.04)
  Week 52: Special Nonverbal Composite (SNC): number analyzed (Participants) | 11 | 26
  Week 52: Special Nonverbal Composite (SNC) | -11.8 (5.38) | -5.0 (3.74)

6. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales, Second Edition (VABS-II) Standard Scores of Other Domains at Weeks 16, 28, 40, 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The standard scores represent a score (mean = 100 and standard deviation of 15) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in adaptive functioning. Communication, daily living skills, socialization and motor skills domains were reported here. The range for individual standard scores is 20-160.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: Communication: number analyzed (Participants) | 15 | 33
  Week 16: Communication | -2.8 (2.65) | -1.7 (1.94)
  Week 16: Daily Living Skills: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills | -3.5 (3.11) | -3.5 (2.33)
  Week 16: Socialization: number analyzed (Participants) | 15 | 32
  Week 16: Socialization | -4.0 (2.43) | -2.0 (2.05)
  Week 16: Motor Skills: number analyzed (Participants) | 12 | 27
  Week 16: Motor Skills | 1.0 (2.00) | 0.0 (1.46)
  Week 28: Communication: number analyzed (Participants) | 15 | 30
  Week 28: Communication | -2.4 (2.80) | -0.3 (2.08)
  Week 28: Daily Living Skills: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills | 0.1 (3.40) | -2.0 (2.53)
  Week 28: Socialization: number analyzed (Participants) | 15 | 30
  Week 28: Socialization | -0.8 (2.37) | -0.2 (2.02)
  Week 28: Motor Skills: number analyzed (Participants) | 12 | 25
  Week 28: Motor Skills | -0.2 (2.46) | 0.7 (1.77)
  Week 40: Communication: number analyzed (Participants) | 14 | 32
  Week 40: Communication | -3.5 (2.82) | -4.6 (2.07)
  Week 40: Daily Living Skills: number analyzed (Participants) | 15 | 31
  Week 40: Daily Living Skills | -2.0 (3.47) | -3.7 (2.57)
  Week 40: Socialization: number analyzed (Participants) | 15 | 32
  Week 40: Socialization | -4.0 (2.65) | -3.8 (2.17)
  Week 40: Motor Skills: number analyzed (Participants) | 12 | 26
  Week 40: Motor Skills | -2.2 (2.47) | -1.1 (1.77)
  Week 52: Communication: number analyzed (Participants) | 15 | 32
  Week 52: Communication | -4.8 (2.99) | -5.8 (2.18)
  Week 52: Daily Living Skills: number analyzed (Participants) | 14 | 32
  Week 52: Daily Living Skills | -4.5 (3.50) | -4.4 (2.57)
  Week 52: Socialization: number analyzed (Participants) | 15 | 32
  Week 52: Socialization | -5.8 (2.72) | -2.8 (2.21)
  Week 52: Motor Skills: number analyzed (Participants) | 12 | 26
  Week 52: Motor Skills | -5.7 (2.47) | -1.3 (1.77)

7. Secondary Outcome: Change From Baseline of Age Equivalent Score for Early Years of Core Subtests of the Differential Ability Scales, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The early years battery is designed for children ages 2 years 6 months through 6 years 11 months. Standardized scores were converted to age equivalent scores to measure ability, skill, and knowledge expressed as the age at which most individuals reach the same level. The mean age equivalent score is obtained by averaging out the age-equivalent scores. The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 32
Score on a scale
  Week 16: Verbal Comprehension: number analyzed (Participants) | 14 | 29
  Week 16: Verbal Comprehension | 0.05 (0.748) | 0.03 (0.700)
  Week 16: Picture Similarities: number analyzed (Participants) | 14 | 29
  Week 16: Picture Similarities | 0.00 (1.056) | 0.48 (1.002)
  Week 16: Naming Vocabulary: number analyzed (Participants) | 14 | 29
  Week 16: Naming Vocabulary | 0.18 (0.432) | -0.02 (0.702)
  Week 16: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 16: Pattern Construction | -0.14 (0.435) | 0.25 (0.475)
  Week 16: Matrices: number analyzed (Participants) | 10 | 27
  Week 16: Matrices | 0.48 (2.076) | 0.38 (1.322)
  Week 16: Copying: number analyzed (Participants) | 10 | 27
  Week 16: Copying | 0.05 (0.197) | 0.10 (0.211)
  Week 28: Verbal Comprehension: number analyzed (Participants) | 11 | 28
  Week 28: Verbal Comprehension | -0.16 (0.846) | 0.39 (0.780)
  Week 28: Picture Similarities: number analyzed (Participants) | 11 | 28
  Week 28: Picture Similarities | 0.39 (1.051) | 0.43 (0.693)
  Week 28: Naming Vocabulary: number analyzed (Participants) | 11 | 28
  Week 28: Naming Vocabulary | 0.27 (0.325) | 0.26 (0.870)
  Week 28: Pattern Construction: number analyzed (Participants) | 11 | 28
  Week 28: Pattern Construction | -0.18 (0.389) | 0.29 (0.543)
  Week 28: Matrices: number analyzed (Participants) | 8 | 25
  Week 28: Matrices | 0.78 (1.089) | 0.51 (1.802)
  Week 28: Copying: number analyzed (Participants) | 8 | 25
  Week 28: Copying | 0.06 (0.291) | 0.14 (0.361)
  Week 40: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 40: Verbal Comprehension | -0.11 (0.783) | 0.17 (0.519)
  Week 40: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 40: Picture Similarities | 0.23 (1.277) | 0.52 (1.081)
  Week 40: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 40: Naming Vocabulary | -0.04 (0.950) | 0.17 (0.721)
  Week 40: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 40: Pattern Construction | -0.02 (0.317) | 0.43 (0.733)
  Week 40: Matrices: number analyzed (Participants) | 10 | 24
  Week 40: Matrices | 0.15 (1.890) | 0.45 (1.721)
  Week 40: Copying: number analyzed (Participants) | 10 | 24
  Week 40: Copying | 0.33 (0.472) | 0.30 (0.556)
  Week 52: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 52: Verbal Comprehension | 0.16 (1.090) | 0.32 (0.657)
  Week 52: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 52: Picture Similarities | 0.27 (1.207) | 0.84 (1.215)
  Week 52: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 52: Naming Vocabulary | 0.16 (0.959) | 0.34 (1.006)
  Week 52: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 52: Pattern Construction | 0.02 (0.360) | 0.31 (0.660)
  Week 52: Matrices: number analyzed (Participants) | 10 | 24
  Week 52: Matrices | 0.00 (1.863) | 0.64 (1.771)
  Week 52: Copying: number analyzed (Participants) | 10 | 23
  Week 52: Copying | 0.20 (0.438) | 0.28 (0.502)

8. Secondary Outcome: Change From Baseline of Age Equivalents for School Age of Core Subtests of the Differential Ability Scales, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The school age battery is designed for children ages 7 years 0 months through 17 years 11 months. Standardized scores were converted to age equivalent scores to measure ability, skill, and knowledge expressed as the age at which most individuals reach the same level. The mean age equivalent score is obtained by averaging out the age-equivalent scores. The higher score indicates greater cognitive ability. The subtest score represents a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability. In the below table, SQR stands for "Sequential & Quantitative Reasoning".
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 1 | 4
Score on a scale
  Week 16: Recall of Designs: number analyzed (Participants) | 1 | 2
  Week 16: Recall of Designs | -1.75 (NA) — Standard deviation was not calculated due to less number of participants. | 1.00 (1.414)
  Week 16: Word Definitions: number analyzed (Participants) | 1 | 2
  Week 16: Word Definitions | 1.50 (NA) — Standard deviation was not calculated due to less number of participants. | 0.25 (0.707)
  Week 16: Pattern Construction: number analyzed (Participants) | 1 | 2
  Week 16: Pattern Construction | 1.00 (NA) — Standard deviation was not calculated due to less number of participants. | -0.13 (0.177)
  Week 16: Matrices: number analyzed (Participants) | 1 | 2
  Week 16: Matrices | -0.75 (NA) — Standard deviation was not calculated due to less number of participants. | 0.38 (2.652)
  Week 16: Verbal Similarities: number analyzed (Participants) | 1 | 2
  Week 16: Verbal Similarities | 0.75 (NA) — Standard deviation was not calculated due to less number of participants. | 0.63 (0.884)
  Week 16: SQR: number analyzed (Participants) | 1 | 2
  Week 16: SQR | 1.17 (NA) — Standard deviation was not calculated due to less number of participants. | 0.63 (0.884)
  Week 28: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 28: Recall of Designs | -1.00 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 28: Word Definitions | 1.50 (NA) — Standard deviation was not calculated due to less number of participants. | -0.25 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 28: Pattern Construction | 1.50 (NA) — Standard deviation was not calculated due to less number of participants. | -1.75 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Matrices: number analyzed (Participants) | 1 | 1
  Week 28: Matrices | -2.50 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 28: Verbal Similarities | 0.75 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: SQR: number analyzed (Participants) | 1 | 1
  Week 28: SQR | 0.25 (NA) — Standard deviation was not calculated due to less number of participants. | 0.75 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 40: Recall of Designs | -2.00 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 40: Word Definitions | 1.50 (NA) — Standard deviation was not calculated due to less number of participants. | -0.25 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 40: Pattern Construction | 1.92 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Matrices: number analyzed (Participants) | 1 | 1
  Week 40: Matrices | -2.25 (NA) — Standard deviation was not calculated due to less number of participants. | 1.25 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 40: Verbal Similarities | 0.75 (NA) — Standard deviation was not calculated due to less number of participants. | 1.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: SQR: number analyzed (Participants) | 1 | 1
  Week 40: SQR | 1.17 (NA) — Standard deviation was not calculated due to less number of participants. | 1.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 52: Recall of Designs | -2.50 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 52: Word Definitions | 1.75 (NA) — Standard deviation was not calculated due to less number of participants. | -0.25 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 52: Pattern Construction | 1.92 (NA) — Standard deviation was not calculated due to less number of participants. | -2.75 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Matrices: number analyzed (Participants) | 1 | 1
  Week 52: Matrices | -0.25 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 52: Verbal Similarities | 1.17 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: SQR: number analyzed (Participants) | 1 | 1
  Week 52: SQR | 0.67 (NA) — Standard deviation was not calculated due to less number of participants. | 1.00 (NA) — Standard deviation was not calculated due to less number of participants.

9. Secondary Outcome: Change From Baseline of Development Quotients for Early Years of Core Subtests of the Differential Ability Scales, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The early years battery is designed for children ages 2 years 6 months through 6 years 11 months. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of chronological age
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 14 | 32
Percentage of chronological age
  Week 16: Verbal Comprehension: number analyzed (Participants) | 14 | 29
  Week 16: Verbal Comprehension | -5.91 (13.454) | -4.71 (12.990)
  Week 16: Picture Similarities: number analyzed (Participants) | 14 | 29
  Week 16: Picture Similarities | -4.91 (16.959) | 3.41 (19.157)
  Week 16: Naming Vocabulary: number analyzed (Participants) | 14 | 29
  Week 16: Naming Vocabulary | -2.09 (7.758) | -5.44 (11.221)
  Week 16: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 16: Pattern Construction | -7.79 (7.339) | -0.43 (9.213)
  Week 16: Matrices: number analyzed (Participants) | 10 | 27
  Week 16: Matrices | 4.60 (30.134) | 0.57 (24.054)
  Week 16: Copying: number analyzed (Participants) | 10 | 27
  Week 16: Copying | -4.59 (4.206) | -4.15 (4.794)
  Week 28: Verbal Comprehension: number analyzed (Participants) | 11 | 28
  Week 28: Verbal Comprehension | -14.05 (16.558) | -1.46 (15.790)
  Week 28: Picture Similarities: number analyzed (Participants) | 11 | 28
  Week 28: Picture Similarities | -1.89 (17.409) | 0.03 (14.733)
  Week 28: Naming Vocabulary: number analyzed (Participants) | 11 | 28
  Week 28: Naming Vocabulary | -3.78 (6.970) | -3.76 (18.235)
  Week 28: Pattern Construction: number analyzed (Participants) | 11 | 28
  Week 28: Pattern Construction | -11.95 (7.039) | -3.09 (10.708)
  Week 28: Matrices: number analyzed (Participants) | 8 | 25
  Week 28: Matrices | 2.96 (18.576) | 0.45 (34.931)
  Week 28: Copying: number analyzed (Participants) | 8 | 25
  Week 28: Copying | -6.88 (5.759) | -6.66 (7.820)
  Week 40: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 40: Verbal Comprehension | -15.40 (17.544) | -8.97 (11.618)
  Week 40: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 40: Picture Similarities | -6.86 (19.775) | -3.11 (20.029)
  Week 40: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 40: Naming Vocabulary | -10.02 (13.307) | -8.96 (14.427)
  Week 40: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 40: Pattern Construction | -11.56 (6.989) | -3.89 (13.394)
  Week 40: Matrices: number analyzed (Participants) | 10 | 24
  Week 40: Matrices | -7.79 (24.750) | -5.73 (32.283)
  Week 40: Copying: number analyzed (Participants) | 10 | 24
  Week 40: Copying | -6.15 (9.533) | -7.69 (11.208)
  Week 52: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 52: Verbal Comprehension | -14.49 (22.614) | -8.59 (13.473)
  Week 52: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 52: Picture Similarities | -8.32 (19.393) | 0.56 (22.325)
  Week 52: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 52: Naming Vocabulary | -10.29 (13.522) | -8.20 (18.543)
  Week 52: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 52: Pattern Construction | -13.59 (8.232) | -8.49 (11.528)
  Week 52: Matrices: number analyzed (Participants) | 10 | 24
  Week 52: Matrices | -12.47 (23.892) | -5.53 (32.584)
  Week 52: Copying: number analyzed (Participants) | 10 | 23
  Week 52: Copying | -10.19 (9.608) | -10.34 (10.429)

10. Secondary Outcome: Change From Baseline of Development Quotients for School Age of Core Subtests of the Differential Ability Scales, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The school age battery is designed for children ages 7 years 0 months through 17 years 11 months. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability. In the below table, SQR stands for "Sequential & Quantitative Reasoning".
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of chronological age
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 1 | 4
Percentage of chronological age
  Week 16: Recall of Designs: number analyzed (Participants) | 1 | 2
  Week 16: Recall of Designs | -15.10 (NA) — Standard deviation was not calculated due to less number of participants. | 9.20 (17.395)
  Week 16: Word Definitions: number analyzed (Participants) | 1 | 2
  Week 16: Word Definitions | 9.60 (NA) — Standard deviation was not calculated due to less number of participants. | 0.00 (9.192)
  Week 16: Pattern Construction: number analyzed (Participants) | 1 | 2
  Week 16: Pattern Construction | 5.70 (NA) — Standard deviation was not calculated due to less number of participants. | -4.85 (2.051)
  Week 16: Matrices: number analyzed (Participants) | 1 | 2
  Week 16: Matrices | -7.60 (NA) — Standard deviation was not calculated due to less number of participants. | 2.40 (33.800)
  Week 16: Verbal Similarities: number analyzed (Participants) | 1 | 2
  Week 16: Verbal Similarities | 3.70 (NA) — Standard deviation was not calculated due to less number of participants. | 4.65 (10.960)
  Week 16: SQR: number analyzed (Participants) | 1 | 2
  Week 16: SQR | 6.70 (NA) — Standard deviation was not calculated due to less number of participants. | 4.50 (10.748)
  Week 28: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 28: Recall of Designs | -10.40 (NA) — Standard deviation was not calculated due to less number of participants. | -4.80 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 28: Word Definitions | 8.70 (NA) — Standard deviation was not calculated due to less number of participants. | -8.20 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 28: Pattern Construction | 8.40 (NA) — Standard deviation was not calculated due to less number of participants. | -26.90 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Matrices: number analyzed (Participants) | 1 | 1
  Week 28: Matrices | -21.40 (NA) — Standard deviation was not calculated due to less number of participants. | -3.40 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 28: Verbal Similarities | 2.60 (NA) — Standard deviation was not calculated due to less number of participants. | -4.80 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: SQR: number analyzed (Participants) | 1 | 1
  Week 28: SQR | -1.20 (NA) — Standard deviation was not calculated due to less number of participants. | 4.40 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 40: Recall of Designs | -18.70 (NA) — Standard deviation was not calculated due to less number of participants. | -6.50 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 40: Word Definitions | 7.50 (NA) — Standard deviation was not calculated due to less number of participants. | -9.90 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 40: Pattern Construction | 10.20 (NA) — Standard deviation was not calculated due to less number of participants. | -7.20 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Matrices: number analyzed (Participants) | 1 | 1
  Week 40: Matrices | -20.50 (NA) — Standard deviation was not calculated due to less number of participants. | 10.40 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 40: Verbal Similarities | 1.40 (NA) — Standard deviation was not calculated due to less number of participants. | 5.50 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: SQR: number analyzed (Participants) | 1 | 1
  Week 40: SQR | 4.20 (NA) — Standard deviation was not calculated due to less number of participants. | 5.50 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 52: Recall of Designs | -22.90 (NA) — Standard deviation was not calculated due to less number of participants. | -8.10 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 52: Word Definitions | 8.40 (NA) — Standard deviation was not calculated due to less number of participants. | -11.50 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 52: Pattern Construction | 9.20 (NA) — Standard deviation was not calculated due to less number of participants. | -41.00 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Matrices: number analyzed (Participants) | 1 | 1
  Week 52: Matrices | -6.90 (NA) — Standard deviation was not calculated due to less number of participants. | -5.70 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 52: Verbal Similarities | 3.40 (NA) — Standard deviation was not calculated due to less number of participants. | -8.10 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: SQR: number analyzed (Participants) | 1 | 1
  Week 52: SQR | -0.40 (NA) — Standard deviation was not calculated due to less number of participants. | 3.60 (NA) — Standard deviation was not calculated due to less number of participants.

11. Secondary Outcome: Change From Baseline of T-scores for Early Years of Core Subtests of the Differential Ability Scale, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The early years battery is designed for children ages 2 years 6 months through 6 years 11 months. The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 14 | 32
T-score
  Week 16: Verbal Comprehension: number analyzed (Participants) | 14 | 29
  Week 16: Verbal Comprehension | -1.7 (7.27) | -3.6 (9.30)
  Week 16: Picture Similarities: number analyzed (Participants) | 14 | 29
  Week 16: Picture Similarities | -2.3 (9.62) | 2.1 (9.10)
  Week 16: Naming Vocabulary: number analyzed (Participants) | 14 | 29
  Week 16: Naming Vocabulary | -0.1 (6.01) | -2.4 (6.21)
  Week 16: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 16: Pattern Construction | -6.4 (6.01) | 0.6 (8.77)
  Week 16: Matrices: number analyzed (Participants) | 10 | 27
  Week 16: Matrices | -4.3 (17.73) | 0.4 (14.65)
  Week 16: Copying: number analyzed (Participants) | 10 | 27
  Week 16: Copying | -2.2 (8.48) | -0.5 (8.76)
  Week 28: Verbal Comprehension: number analyzed (Participants) | 11 | 28
  Week 28: Verbal Comprehension | -2.2 (10.32) | -1.8 (11.33)
  Week 28: Picture Similarities: number analyzed (Participants) | 11 | 28
  Week 28: Picture Similarities | 2.6 (7.97) | 0.3 (6.28)
  Week 28: Naming Vocabulary: number analyzed (Participants) | 11 | 28
  Week 28: Naming Vocabulary | -0.3 (4.13) | -2.0 (7.79)
  Week 28: Pattern Construction: number analyzed (Participants) | 11 | 28
  Week 28: Pattern Construction | -8.9 (5.36) | -1.5 (9.74)
  Week 28: Matrices: number analyzed (Participants) | 8 | 25
  Week 28: Matrices | 2.9 (6.47) | 0.6 (16.09)
  Week 28: Copying: number analyzed (Participants) | 8 | 25
  Week 28: Copying | -0.9 (6.36) | -1.6 (11.26)
  Week 40: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 40: Verbal Comprehension | -4.9 (8.21) | -3.4 (6.55)
  Week 40: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 40: Picture Similarities | 0.1 (13.04) | -2.0 (9.81)
  Week 40: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 40: Naming Vocabulary | -4.4 (9.69) | -3.9 (7.54)
  Week 40: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 40: Pattern Construction | -8.7 (5.78) | -2.6 (11.24)
  Week 40: Matrices: number analyzed (Participants) | 10 | 24
  Week 40: Matrices | -7.4 (16.87) | -3.2 (16.71)
  Week 40: Copying: number analyzed (Participants) | 10 | 24
  Week 40: Copying | -1.8 (11.39) | -0.1 (12.69)
  Week 52: Verbal Comprehension: number analyzed (Participants) | 14 | 27
  Week 52: Verbal Comprehension | -4.6 (11.21) | -4.9 (11.10)
  Week 52: Picture Similarities: number analyzed (Participants) | 14 | 27
  Week 52: Picture Similarities | -1.7 (15.41) | 0.3 (10.44)
  Week 52: Naming Vocabulary: number analyzed (Participants) | 14 | 27
  Week 52: Naming Vocabulary | -2.7 (8.59) | -3.2 (8.54)
  Week 52: Pattern Construction: number analyzed (Participants) | 14 | 27
  Week 52: Pattern Construction | -10.9 (8.03) | -6.1 (10.90)
  Week 52: Matrices: number analyzed (Participants) | 10 | 24
  Week 52: Matrices | -8.5 (15.52) | -0.8 (17.00)
  Week 52: Copying: number analyzed (Participants) | 10 | 23
  Week 52: Copying | -4.0 (10.68) | -2.4 (12.07)

12. Secondary Outcome: Change From Baseline of T-scores for School Age of Core Subtests of the Differential Ability Scale, Second Edition (DAS-II) at Weeks 16, 28, 40 and 52
Description: The DAS-II was used to assess cognitive development in all randomized participants. The school age battery is designed for children ages 7 years 0 months through 17 years 11 months. The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability. In the below table, SQR stands for "Sequential & Quantitative Reasoning".
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 1 | 4
Score on a scale
  Week 16: Recall of Designs: number analyzed (Participants) | 1 | 2
  Week 16: Recall of Designs | -10.0 (NA) — Standard deviation was not calculated due to less number of participants. | 5.0 (12.73)
  Week 16: Word Definitions: number analyzed (Participants) | 1 | 2
  Week 16: Word Definitions | 7.0 (NA) — Standard deviation was not calculated due to less number of participants. | -0.5 (7.78)
  Week 16: Pattern Construction: number analyzed (Participants) | 1 | 2
  Week 16: Pattern Construction | 3.0 (NA) — Standard deviation was not calculated due to less number of participants. | -2.0 (1.41)
  Week 16: Matrices: number analyzed (Participants) | 1 | 2
  Week 16: Matrices | -5.0 (NA) — Standard deviation was not calculated due to less number of participants. | -0.5 (12.02)
  Week 16: Verbal Similarities: number analyzed (Participants) | 1 | 2
  Week 16: Verbal Similarities | 4.0 (NA) — Standard deviation was not calculated due to less number of participants. | -4.0 (8.49)
  Week 16: SQR: number analyzed (Participants) | 1 | 2
  Week 16: SQR | 2.0 (NA) — Standard deviation was not calculated due to less number of participants. | 3.0 (2.83)
  Week 28: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 28: Recall of Designs | -7.0 (NA) — Standard deviation was not calculated due to less number of participants. | 10.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 28: Word Definitions | 5.0 (NA) — Standard deviation was not calculated due to less number of participants. | -8.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 28: Pattern Construction | 4.0 (NA) — Standard deviation was not calculated due to less number of participants. | -19.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Matrices: number analyzed (Participants) | 1 | 1
  Week 28: Matrices | -12.0 (NA) — Standard deviation was not calculated due to less number of participants. | -9.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 28: Verbal Similarities | 3.0 (NA) — Standard deviation was not calculated due to less number of participants. | -10.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 28: SQR: number analyzed (Participants) | 1 | 1
  Week 28: SQR | -2.0 (NA) — Standard deviation was not calculated due to less number of participants. | 9.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 40: Recall of Designs | -14.0 (NA) — Standard deviation was not calculated due to less number of participants. | -4.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 40: Word Definitions | 5.0 (NA) — Standard deviation was not calculated due to less number of participants. | -16.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 40: Pattern Construction | 5.0 (NA) — Standard deviation was not calculated due to less number of participants. | -3.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Matrices: number analyzed (Participants) | 1 | 1
  Week 40: Matrices | -11.0 (NA) — Standard deviation was not calculated due to less number of participants. | 1.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 40: Verbal Similarities | 2.0 (NA) — Standard deviation was not calculated due to less number of participants. | 1.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 40: SQR: number analyzed (Participants) | 1 | 1
  Week 40: SQR | 1.0 (NA) — Standard deviation was not calculated due to less number of participants. | 10.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Recall of Designs: number analyzed (Participants) | 1 | 1
  Week 52: Recall of Designs | -17.0 (NA) — Standard deviation was not calculated due to less number of participants. | -4.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Word Definitions: number analyzed (Participants) | 1 | 1
  Week 52: Word Definitions | 6.0 (NA) — Standard deviation was not calculated due to less number of participants. | -17.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Pattern Construction: number analyzed (Participants) | 1 | 1
  Week 52: Pattern Construction | 4.0 (NA) — Standard deviation was not calculated due to less number of participants. | -30.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Matrices: number analyzed (Participants) | 1 | 1
  Week 52: Matrices | -4.0 (NA) — Standard deviation was not calculated due to less number of participants. | -5.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: Verbal Similarities: number analyzed (Participants) | 1 | 1
  Week 52: Verbal Similarities | 5.0 (NA) — Standard deviation was not calculated due to less number of participants. | -10.0 (NA) — Standard deviation was not calculated due to less number of participants.
  Week 52: SQR | -2.0 (NA) — Standard deviation was not calculated due to less number of participants. | 9.0 (NA) — Standard deviation was not calculated due to less number of participants.

13. Secondary Outcome: Change From Baseline of Age Equivalents Scores of Sub-domains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at Weeks 16, 28, 40 and 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. Standardized scores (range 40-160) were converted to age equivalent scores to measure ability, skill, and knowledge expressed as the age at which most individuals reach the same level. The mean age equivalent score is obtained by averaging out the age-equivalent scores for the all the sub-domains except for Gross and Fine motor skills (range: 0, unbound). A positive value indicates improvement in health and cognition.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: Communication- Expressive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Expressive | 0.09 (0.512) | 0.12 (0.544)
  Week 16: Communication- Receptive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Receptive | -0.09 (1.020) | -0.32 (1.845)
  Week 16: Communication- Written: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Written | 0.08 (0.406) | 0.02 (0.572)
  Week 16: Daily Living Skills- Community: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Community | 0.16 (0.583) | 0.05 (0.710)
  Week 16: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Domestic | 0.02 (1.477) | -0.09 (1.149)
  Week 16: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Personal | -0.23 (0.864) | -0.11 (0.599)
  Week 16: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 16: Socialization- Coping Skills | -0.16 (0.712) | -0.09 (0.792)
  Week 16: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Interpersonal Relationship | -0.09 (0.749) | 0.04 (0.637)
  Week 16: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Play and Leisure Time | 0.21 (0.934) | 0.11 (0.783)
  Week 16: Motor Skills- Fine: number analyzed (Participants) | 12 | 27
  Week 16: Motor Skills- Fine | 0.30 (0.499) | 0.29 (0.429)
  Week 16: Motor Skills- Gross: number analyzed (Participants) | 12 | 28
  Week 16: Motor Skills- Gross | 0.17 (0.607) | 0.36 (0.736)
  Week 28: Communication- Expressive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Expressive | 0.28 (0.669) | 0.36 (0.806)
  Week 28: Communication- Receptive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Receptive | 0.83 (2.393) | 0.44 (1.333)
  Week 28: Communication- Written: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Written | 0.21 (0.663) | 0.18 (0.525)
  Week 28: Daily Living Skills- Community: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Community | 0.22 (0.701) | 0.26 (0.762)
  Week 28: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Domestic | 0.67 (1.481) | 0.34 (1.326)
  Week 28: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Personal | 0.48 (1.260) | 0.16 (0.544)
  Week 28: Socialization- Coping Skills: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Coping Skills | 0.29 (0.731) | 0.27 (0.982)
  Week 28: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Interpersonal Relationship | 0.07 (0.884) | 0.43 (0.876)
  Week 28: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Play and Leisure Time | 0.62 (0.818) | 0.51 (1.017)
  Week 28: Motor Skills- Fine: number analyzed (Participants) | 12 | 25
  Week 28: Motor Skills- Fine | 0.30 (0.403) | 0.37 (0.533)
  Week 28: Motor Skills- Gross: number analyzed (Participants) | 12 | 26
  Week 28: Motor Skills- Gross | 0.41 (0.588) | 0.82 (1.061)
  Week 40: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Expressive | 0.28 (0.679) | 0.30 (0.764)
  Week 40: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Receptive | 0.80 (2.388) | -0.07 (2.015)
  Week 40: Communication- Written: number analyzed (Participants) | 14 | 32
  Week 40: Communication- Written | 0.30 (0.699) | 0.00 (0.740)
  Week 40: Daily Living Skills- Community: number analyzed (Participants) | 15 | 31
  Week 40: Daily Living Skills- Community | 0.38 (0.640) | 0.02 (0.760)
  Week 40: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Domestic | 0.72 (1.542) | 0.39 (1.420)
  Week 40: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Personal | 0.18 (0.720) | 0.29 (0.587)
  Week 40: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Coping Skills | 0.14 (1.178) | 0.26 (1.581)
  Week 40: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Interpersonal Relationship | 0.05 (0.796) | 0.10 (0.973)
  Week 40: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Play and Leisure Time | 0.44 (0.808) | 0.31 (0.921)
  Week 40: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 40: Motor Skills- Fine | 0.44 (0.453) | 0.44 (0.640)
  Week 40: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 40: Motor Skills- Gross | 0.33 (0.662) | 0.73 (0.990)
  Week 52: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Expressive | 0.32 (0.973) | 0.34 (0.858)
  Week 52: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Receptive | 1.25 (2.253) | -0.05 (1.953)
  Week 52: Communication- Written: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Written | 0.16 (0.485) | 0.11 (0.783)
  Week 52: Daily Living Skills- Community: number analyzed (Participants) | 14 | 32
  Week 52: Daily Living Skills- Community | 0.36 (0.603) | 0.30 (0.941)
  Week 52: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Domestic | 0.27 (1.678) | 0.37 (1.405)
  Week 52: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Personal | 0.42 (0.572) | 0.35 (0.840)
  Week 52: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Coping Skills | 0.29 (1.211) | 0.31 (1.189)
  Week 52: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Interpersonal Relationship | 0.00 (0.752) | 0.36 (1.005)
  Week 52: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Play and Leisure Time | 0.67 (1.446) | 0.45 (0.839)
  Week 52: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 52: Motor Skills- Fine | 0.38 (0.365) | 0.58 (0.645)
  Week 52: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 52: Motor Skills- Gross | 0.25 (0.773) | 0.93 (1.008)

14. Secondary Outcome: Change From Baseline of Development Quotients of Sub-domains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at Weeks 16, 28, 40 and 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The DQ is a means to express a neurodevelopmental/cognitive delay. The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0, 100). The overall DQ score is calculated from the mean age-equivalent score obtained by averaging out the age equivalent scores for the all the sub-domains except for Gross and Fine motor skills. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). A positive value indicates improvement in health and cognition.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage of chronological age
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Percentage of chronological age
  Week 16: Communication- Expressive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Expressive | -1.09 (7.866) | -2.57 (11.781)
  Week 16: Communication- Receptive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Receptive | -2.58 (14.735) | -8.19 (26.774)
  Week 16: Communication- Written: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Written | -4.10 (8.727) | -5.62 (12.554)
  Week 16: Daily Living Skills- Community: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Community | -0.37 (12.814) | -4.48 (15.498)
  Week 16: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Domestic | -2.80 (30.338) | -7.18 (24.610)
  Week 16: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Personal | -9.94 (21.052) | -6.35 (11.185)
  Week 16: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 16: Socialization- Coping Skills | -9.08 (14.414) | -6.56 (15.923)
  Week 16: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Interpersonal Relationship | -3.87 (9.602) | -3.17 (14.610)
  Week 16: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Play and Leisure Time | 1.66 (18.903) | -0.64 (15.366)
  Week 16: Motor Skills- Fine: number analyzed (Participants) | 12 | 27
  Week 16: Motor Skills- Fine | 0.48 (12.969) | 0.00 (10.308)
  Week 16: Motor Skills- Gross: number analyzed (Participants) | 12 | 28
  Week 16: Motor Skills- Gross | -3.92 (15.524) | 1.28 (15.410)
  Week 28: Communication- Expressive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Expressive | -0.23 (11.301) | -0.59 (14.480)
  Week 28: Communication- Receptive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Receptive | 3.30 (24.423) | 0.50 (17.058)
  Week 28: Communication- Written: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Written | -5.15 (13.510) | -6.54 (11.339)
  Week 28: Daily Living Skills- Community: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Community | -3.07 (13.984) | -2.80 (15.937)
  Week 28: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Domestic | 6.75 (28.703) | -3.37 (25.635)
  Week 28: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Personal | 3.41 (26.699) | -4.27 (12.124)
  Week 28: Socialization- Coping Skills: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Coping Skills | -4.88 (15.881) | -2.45 (19.142)
  Week 28: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Interpersonal Relationship | -2.30 (13.889) | 2.16 (17.844)
  Week 28: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Play and Leisure Time | 8.17 (17.767) | 4.49 (20.413)
  Week 28: Motor Skills- Fine: number analyzed (Participants) | 12 | 25
  Week 28: Motor Skills- Fine | -2.86 (9.014) | -2.05 (12.124)
  Week 28: Motor Skills- Gross: number analyzed (Participants) | 12 | 26
  Week 28: Motor Skills- Gross | -3.05 (15.068) | 7.78 (21.604)
  Week 40: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Expressive | -2.35 (10.521) | -3.74 (12.846)
  Week 40: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Receptive | 0.31 (22.511) | -8.32 (29.716)
  Week 40: Communication- Written: number analyzed (Participants) | 14 | 32
  Week 40: Communication- Written | -5.39 (14.066) | -13.31 (15.173)
  Week 40: Daily Living Skills- Community: number analyzed (Participants) | 15 | 31
  Week 40: Daily Living Skills- Community | -2.29 (13.856) | -9.72 (15.988)
  Week 40: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Domestic | 4.40 (27.464) | -4.53 (27.189)
  Week 40: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Personal | -5.54 (14.516) | -4.33 (11.630)
  Week 40: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Coping Skills | -11.75 (18.650) | -7.31 (22.758)
  Week 40: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Interpersonal Relationship | -5.47 (13.597) | -6.38 (18.307)
  Week 40: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Play and Leisure Time | 1.83 (18.194) | -1.20 (19.009)
  Week 40: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 40: Motor Skills- Fine | -3.51 (10.891) | -4.04 (14.407)
  Week 40: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 40: Motor Skills- Gross | -9.01 (18.404) | 1.75 (18.235)
  Week 52: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Expressive | -4.87 (13.094) | -5.22 (14.616)
  Week 52: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Receptive | 5.58 (18.225) | -10.14 (29.190)
  Week 52: Communication- Written: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Written | -11.22 (10.973) | -13.90 (16.079)
  Week 52: Daily Living Skills- Community: number analyzed (Participants) | 14 | 32
  Week 52: Daily Living Skills- Community | -6.46 (13.154) | -7.10 (18.149)
  Week 52: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Domestic | -6.81 (28.704) | -8.64 (27.817)
  Week 52: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Personal | -3.64 (11.626) | -5.79 (15.032)
  Week 52: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Coping Skills | -11.26 (19.505) | -6.54 (20.142)
  Week 52: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Interpersonal Relationship | -8.53 (12.960) | -4.46 (17.892)
  Week 52: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Play and Leisure Time | 1.95 (25.499) | -0.83 (15.499)
  Week 52: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 52: Motor Skills- Fine | -8.58 (8.790) | -4.67 (15.370)
  Week 52: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 52: Motor Skills- Gross | -14.54 (21.617) | 2.46 (18.655)

15. Secondary Outcome: Change From Baseline of V-Scale Scores of Sub-domains of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at Weeks 16, 28, 40 and 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (a composite of the other 4 domains). The V-scale scores represent a score (mean = 15 and standard deviation of 3; range: 1-24) on which higher scores indicate a higher level of adaptive functioning. A positive change value indicates improvement in adaptive functioning.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: Communication- Expressive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Expressive | -0.1 (1.81) | -0.4 (2.05)
  Week 16: Communication- Receptive: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Receptive | -0.3 (1.84) | -0.7 (1.85)
  Week 16: Communication- Written: number analyzed (Participants) | 15 | 33
  Week 16: Communication- Written | -0.7 (1.83) | -1.1 (2.87)
  Week 16: Daily Living Skills- Community: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Community | -0.3 (1.28) | -0.7 (2.05)
  Week 16: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Domestic | -0.3 (2.61) | -0.7 (1.93)
  Week 16: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 33
  Week 16: Daily Living Skills- Personal | -1.2 (3.23) | -1.2 (2.34)
  Week 16: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 16: Socialization- Coping Skills | -0.6 (1.80) | -0.4 (1.46)
  Week 16: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Interpersonal Relationship | -0.5 (1.46) | -0.3 (1.55)
  Week 16: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 33
  Week 16: Socialization- Play and Leisure Time | 0.2 (2.37) | -0.4 (1.62)
  Week 16: Motor Skills- Fine: number analyzed (Participants) | 12 | 27
  Week 16: Motor Skills- Fine | 0.3 (1.36) | -0.1 (1.33)
  Week 16: Motor Skills- Gross: number analyzed (Participants) | 12 | 28
  Week 16: Motor Skills- Gross | -0.3 (1.61) | 0.0 (2.00)
  Week 28: Communication- Expressive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Expressive | 0.0 (2.00) | -0.3 (2.20)
  Week 28: Communication- Receptive: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Receptive | -0.1 (2.40) | -0.1 (1.17)
  Week 28: Communication- Written: number analyzed (Participants) | 15 | 30
  Week 28: Communication- Written | -0.6 (2.41) | -1.2 (2.04)
  Week 28: Daily Living Skills- Community: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Community | -0.7 (1.75) | -0.7 (1.95)
  Week 28: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Domestic | 0.4 (2.75) | -0.4 (2.11)
  Week 28: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 30
  Week 28: Daily Living Skills- Personal | 0.6 (3.50) | -0.6 (2.21)
  Week 28: Socialization- Coping Skills: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Coping Skills | 0.1 (1.51) | -0.2 (1.43)
  Week 28: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Interpersonal Relationship | -0.4 (1.84) | 0.1 (1.49)
  Week 28: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 30
  Week 28: Socialization- Play and Leisure Time | 1.1 (2.03) | 0.2 (2.04)
  Week 28: Motor Skills- Fine: number analyzed (Participants) | 12 | 25
  Week 28: Motor Skills- Fine | -0.3 (1.06) | -0.3 (1.62)
  Week 28: Motor Skills- Gross: number analyzed (Participants) | 12 | 26
  Week 28: Motor Skills- Gross | -0.2 (2.33) | 0.5 (2.06)
  Week 40: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Expressive | 0.0 (1.85) | -0.8 (1.76)
  Week 40: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 40: Communication- Receptive | -0.2 (2.08) | -0.7 (2.07)
  Week 40: Communication- Written: number analyzed (Participants) | 14 | 32
  Week 40: Communication- Written | -0.9 (2.59) | -2.6 (3.05)
  Week 40: Daily Living Skills- Community: number analyzed (Participants) | 15 | 31
  Week 40: Daily Living Skills- Community | -0.6 (1.59) | -1.6 (1.91)
  Week 40: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Domestic | 0.3 (2.72) | -0.7 (2.66)
  Week 40: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 40: Daily Living Skills- Personal | -0.6 (2.69) | -0.5 (2.09)
  Week 40: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Coping Skills | -0.6 (1.96) | -0.8 (1.80)
  Week 40: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Interpersonal Relationship | -0.8 (1.70) | -0.9 (1.72)
  Week 40: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 40: Socialization- Play and Leisure Time | 0.5 (2.10) | -0.4 (2.24)
  Week 40: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 40: Motor Skills- Fine | -0.3 (1.56) | -0.5 (1.79)
  Week 40: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 40: Motor Skills- Gross | -0.8 (1.90) | -0.1 (2.23)
  Week 52: Communication- Expressive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Expressive | -0.5 (1.88) | -1.0 (2.44)
  Week 52: Communication- Receptive: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Receptive | 0.1 (2.00) | -0.9 (2.08)
  Week 52: Communication- Written: number analyzed (Participants) | 15 | 32
  Week 52: Communication- Written | -2.1 (2.09) | -3.0 (3.25)
  Week 52: Daily Living Skills- Community: number analyzed (Participants) | 14 | 32
  Week 52: Daily Living Skills- Community | -1.5 (1.70) | -1.6 (2.46)
  Week 52: Daily Living Skills- Domestic: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Domestic | -0.5 (2.77) | -0.7 (2.40)
  Week 52: Daily Living Skills- Personal: number analyzed (Participants) | 15 | 32
  Week 52: Daily Living Skills- Personal | -0.1 (1.85) | -0.9 (2.76)
  Week 52: Socialization- Coping Skills: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Coping Skills | -0.7 (1.80) | -0.5 (1.55)
  Week 52: Socialization- Interpersonal Relationship: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Interpersonal Relationship | -1.0 (1.65) | -0.6 (1.81)
  Week 52: Socialization- Play and Leisure Time: number analyzed (Participants) | 15 | 32
  Week 52: Socialization- Play and Leisure Time | -0.1 (3.38) | -0.4 (2.00)
  Week 52: Motor Skills- Fine: number analyzed (Participants) | 12 | 26
  Week 52: Motor Skills- Fine | -1.1 (1.08) | -0.6 (2.06)
  Week 52: Motor Skills- Gross: number analyzed (Participants) | 12 | 27
  Week 52: Motor Skills- Gross | -1.5 (2.07) | -0.1 (2.35)

16. Secondary Outcome: Change From Baseline of V-Scale Scores of Maladaptive Behavior Index and Its Sub-scales at Weeks 16, 28, 40 and 52
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. Maladaptive behavior index is a composite of the internalizing, externalizing, and other types of undesirable behavior that may interfere with the individual's adaptive functioning. The V-scale scores represent a score (mean = 15 and standard deviation of 3; range: 1-24) on which higher scores indicate greater maladaptive behaviors. A positive change value indicates increase of maladaptive behavior.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Score on a scale
  Week 16: Maladaptive Behavior Index: number analyzed (Participants) | 12 | 31
  Week 16: Maladaptive Behavior Index | 0.3 (1.14) | -0.2 (1.18)
  Week 16: Maladaptive Behavior Index- Internalizing: number analyzed (Participants) | 14 | 32
  Week 16: Maladaptive Behavior Index- Internalizing | 0.1 (2.37) | -0.3 (2.31)
  Week 16: Maladaptive Behavior Index- Externalizing: number analyzed (Participants) | 13 | 31
  Week 16: Maladaptive Behavior Index- Externalizing | 0.5 (1.71) | 0.0 (1.53)
  Week 28: Maladaptive Behavior Index: number analyzed (Participants) | 14 | 28
  Week 28: Maladaptive Behavior Index | 0.3 (0.91) | -0.3 (1.27)
  Week 28: Maladaptive Behavior Index- Internalizing: number analyzed (Participants) | 14 | 29
  Week 28: Maladaptive Behavior Index- Internalizing | -0.4 (1.60) | -0.8 (2.11)
  Week 28: Maladaptive Behavior Index- Externalizing: number analyzed (Participants) | 14 | 28
  Week 28: Maladaptive Behavior Index- Externalizing | 0.6 (1.34) | -0.1 (2.01)
  Week 40: Maladaptive Behavior Index: number analyzed (Participants) | 14 | 31
  Week 40: Maladaptive Behavior Index | -0.5 (1.40) | -0.3 (1.13)
  Week 40: Maladaptive Behavior Index- Internalizing: number analyzed (Participants) | 14 | 31
  Week 40: Maladaptive Behavior Index- Internalizing | -1.0 (2.57) | -0.7 (2.98)
  Week 40: Maladaptive Behavior Index- Externalizing: number analyzed (Participants) | 14 | 31
  Week 40: Maladaptive Behavior Index- Externalizing | -0.1 (1.64) | -0.1 (1.29)
  Week 52: Maladaptive Behavior Index: number analyzed (Participants) | 14 | 31
  Week 52: Maladaptive Behavior Index | -0.5 (1.45) | -0.5 (1.41)
  Week 52: Maladaptive Behavior Index- Internalizing: number analyzed (Participants) | 14 | 31
  Week 52: Maladaptive Behavior Index- Internalizing | -1.1 (1.96) | -0.9 (2.72)
  Week 52: Maladaptive Behavior Index- Externalizing: number analyzed (Participants) | 14 | 31
  Week 52: Maladaptive Behavior Index- Externalizing | -0.4 (2.27) | -0.2 (1.69)

17. Secondary Outcome: Observed Maladaptive Levels of Maladaptive Behavior Index and Its Sub-scales of Vineland Adaptive Behavior Scales, Second Edition (VABS-II)
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. Maladaptive behavior index (MBI) is a composite of the internalizing, externalizing, and other types of undesirable behavior that may interfere with the individual's adaptive functioning. The V scale scores represent a score (mean = 15 and standard deviation of 3; range: 1-24) on which higher scores indicate greater maladaptive behaviors. The v-scale score ranges for MBI, externalizing and internalizing scores are defined as clinically significant: 21-24, elevated: 18-20, average: 1-17.
Time Frame: Baseline, Week 16, Week 28, Week 40 and Week 52
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Participants
  Baseline: MBI- Average | 7 | 8
  Baseline: MBI- Elevated | 5 | 20
  Baseline: MBI- Clinically Significant | 2 | 5
  Baseline: Internalizing- Average | 7 | 15
  Baseline: Internalizing- Elevated | 4 | 11
  Baseline: Internalizing- Clinically Significant | 3 | 7
  Baseline: Externalizing- Average | 8 | 11
  Baseline: Externalizing- Elevated | 5 | 19
  Baseline: Externalizing- Clinically Significant | 1 | 3
  Week 16: MBI- Average | 4 | 9
  Week 16: MBI- Elevated | 8 | 17
  Week 16: MBI- Clinically Significant | 1 | 6
  Week 16: Internalizing- Average | 7 | 19
  Week 16: Internalizing- Elevated | 6 | 9
  Week 16: Internalizing- Clinically Significant | 2 | 5
  Week 16: Externalizing- Average | 7 | 13
  Week 16: Externalizing- Elevated | 7 | 14
  Week 16: Externalizing- Clinically Significant | 0 | 5
  Week 28: MBI- Average | 7 | 8
  Week 28: MBI- Elevated | 7 | 16
  Week 28: MBI- Clinically Significant | 1 | 5
  Week 28: Internalizing- Average | 9 | 18
  Week 28: Internalizing- Elevated | 6 | 10
  Week 28: Internalizing- Clinically Significant | 0 | 2
  Week 28: Externalizing- Average | 10 | 11
  Week 28: Externalizing- Elevated | 5 | 14
  Week 28: Externalizing- Clinically Significant | 0 | 4
  Week 40: MBI- Average | 7 | 7
  Week 40: MBI- Elevated | 8 | 21
  Week 40: MBI- Clinically Significant | 0 | 4
  Week 40: Internalizing- Average | 9 | 20
  Week 40: Internalizing- Elevated | 6 | 10
  Week 40: Internalizing- Clinically Significant | 0 | 2
  Week 40: Externalizing- Average | 9 | 12
  Week 40: Externalizing- Elevated | 6 | 18
  Week 40: Externalizing- Clinically Significant | 0 | 2
  Week 52: MBI- Average | 9 | 10
  Week 52: MBI- Elevated | 6 | 18
  Week 52: MBI- Clinically Significant | 0 | 4
  Week 52: Internalizing- Average | 11 | 20
  Week 52: Internalizing- Elevated | 4 | 9
  Week 52: Internalizing- Clinically Significant | 0 | 3
  Week 52: Externalizing- Average | 10 | 15
  Week 52: Externalizing- Elevated | 5 | 15
  Week 52: Externalizing- Clinically Significant | 0 | 2

18. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) of Idursulfase After IT Administration
Description: The Cmax of idursulfase after IT administration was reported.
Time Frame: Pre-dose, 30, 60, 120 minutes, 4, 6, 8, 12, 24, 30 and 36 hour (h) post-dose on Weeks 4, 24, and 48
Population: Pharmacokinetic (PK) population included all participants who received investigational product and participated in the scheduled PK studies, and for whom at least 1 post-dose PK blood sample was collected. PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | IT Treatment
Number analyzed (Participants) | 24
Nanogram per milliliter (ng/mL)
  Week 4 | 253.44 (686.569)
  Week 24: number analyzed (Participants) | 22
  Week 24 | 132.87 (147.044)
  Week 48: number analyzed (Participants) | 22
  Week 48 | 136.15 (127.524)

19. Secondary Outcome: Time to Reach Maximum Drug Concentration (Tmax) of Idursulfase After IT Administration
Description: The tmax of idursulfase after IT administration was reported.
Time Frame: Pre-dose, 30, 60, 120 minutes, 4, 6, 8, 12, 24, 30 and 36 hour (h) post-dose on Weeks 4, 24, and 48
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | IT Treatment
Number analyzed (Participants) | 24
Hour (h)
  Week 4 | 10.07 (7.217)
  Week 24: number analyzed (Participants) | 22
  Week 24 | 10.37 (7.302)
  Week 48: number analyzed (Participants) | 22
  Week 48 | 10.18 (6.609)

20. Secondary Outcome: Area Under the Concentration Versus Time Curve From Zero From the Time of Dosing to the Last Measurable Concentration (AUC0-t) of Idursulfase After IT Administration
Description: The AUC0-t of idursulfase after IT administration was reported.
Time Frame: Pre-dose, 30, 60, 120 minutes, 4, 6, 8, 12, 24, 30 and 36 hour (h) post-dose on Weeks 4, 24, and 48
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | IT Treatment
Number analyzed (Participants) | 24
Nanogram*hour per milliliter (ng*h/mL)
  Week 4 | 2601 (5028.0)
  Week 24: number analyzed (Participants) | 22
  Week 24 | 2949 (4500.4)
  Week 48: number analyzed (Participants) | 22
  Week 48 | 2863 (3571.6)

21. Secondary Outcome: Terminal Half-life (t1/2) of Idursulfase After IT Administration
Description: The t1/2 of idursulfase after IT administration was reported.
Time Frame: Pre-dose, 30, 60, 120 minutes, 4, 6, 8, 12, 24, 30 and 36 hour (h) post-dose on Weeks 4, 24, and 48
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | IT Treatment
Number analyzed (Participants) | 24
Hour (h)
  Week 4: number analyzed (Participants) | 11
  Week 4 | 11.39 (4.996)
  Week 24: number analyzed (Participants) | 12
  Week 24 | 10.68 (2.851)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 11.52 (4.243)

22. Secondary Outcome: Total Body Clearance for Extravascular Administration Divided by the Fraction of Dose Absorbed (CL/F) of Idursulfase After IT Administration
Description: The CL/F of idursulfase after IT administration was reported.
Time Frame: Pre-dose, 30, 60, 120 minutes, 4, 6, 8, 12, 24, 30 and 36 hour (h) post-dose on Weeks 4, 24, and 48
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | IT Treatment
Number analyzed (Participants) | 24
Liter per hour (L/h)
  Week 4: number analyzed (Participants) | 11
  Week 4 | 4.82 (1.753)
  Week 24: number analyzed (Participants) | 12
  Week 24 | 4.54 (2.029)
  Week 48: number analyzed (Participants) | 11
  Week 48 | 3.94 (1.461)

23. Secondary Outcome: Change From Baseline in the Concentration of Glycosaminoglycans (GAG) in Cerebrospinal Fluid (CSF) at Week 52
Description: Change from baseline in the concentration of GAG in CSF was reported.
Time Frame: Baseline, Week 52
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 14 | 30
Nanogram per milliliter (ng/mL) | -124.6 (905.08) | -961.8 (797.01)

24. Secondary Outcome: Concentration of Idursulfase in Cerebrospinal Fluid (CSF)
Description: CSF samples were collected via the IDDD or lumbar puncture prior to the injection of Idursulfase-IT.
Time Frame: Pre-dose on Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48
Population: PK population with number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IT Treatment
Number analyzed (Participants) | 33
ng/mL
  Week 4: number analyzed (Participants) | 31
  Week 4 | 0 (0)
  Week 8: number analyzed (Participants) | 29
  Week 8 | 552.75 (2638.000)
  Week 12: number analyzed (Participants) | 27
  Week 12 | 520.29 (2096.512)
  Week 16: number analyzed (Participants) | 27
  Week 16 | 176.87 (572.459)
  Week 20: number analyzed (Participants) | 29
  Week 20 | 146.66 (553.354)
  Week 24: number analyzed (Participants) | 29
  Week 24 | 268.72 (979.733)
  Week 28: number analyzed (Participants) | 28
  Week 28 | 1471.61 (5893.839)
  Week 32: number analyzed (Participants) | 28
  Week 32 | 141.16 (443.484)
  Week 36: number analyzed (Participants) | 29
  Week 36 | 521.63 (1524.740)
  Week 40: number analyzed (Participants) | 29
  Week 40 | 14436.70 (75712.900)
  Week 44: number analyzed (Participants) | 29
  Week 44 | 1105.46 (5331.560)
  Week 48: number analyzed (Participants) | 27
  Week 48 | 678.50 (3266.592)

25. Secondary Outcome: Participant Response to Quality of Life EuroQol-5D (EQ-5D) Questionnaire at Week 52
Description: The EQ-5D provides a descriptive profile and index value for health status. The questionnaire measures 5 dimensions of health status: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each dimension, there are 5 levels of response: no problems, slight problems, moderate problems, severe problems, and unable to do/extreme problems.
Time Frame: Week 52
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 34
Participants
  Mobility: No problems | 9 | 22
  Mobility: Slight problems | 4 | 7
  Mobility: Moderate problems | 1 | 1
  Mobility: Severe problems | 0 | 0
  Mobility: Unable to do | 0 | 0
  Mobility: Data missing | 1 | 4
  Self-care: No problems | 3 | 6
  Self-care: Slight problems | 4 | 10
  Self-care: Moderate problems | 4 | 7
  Self-care: Severe problems | 0 | 3
  Self-care: Unable to do | 3 | 4
  Self-care: Data missing | 1 | 4
  Usual activities: No problems | 8 | 17
  Usual activities: Slight problems | 3 | 5
  Usual activities: Moderate problems | 2 | 6
  Usual activities: Severe problems | 0 | 1
  Usual activities: Unable to do | 1 | 1
  Usual activities: Data missing | 1 | 4
  Pain/discomfort: No problems | 6 | 20
  Pain/discomfort: Slight problems | 8 | 7
  Pain/discomfort: Moderate problems | 0 | 3
  Pain/discomfort: Severe problems | 0 | 0
  Pain/discomfort: Extreme problems | 0 | 0
  Pain/discomfort: Data missing | 1 | 4
  Anxiety/depression: No problems | 11 | 22
  Anxiety/depression: Slight problems | 3 | 6
  Anxiety/depression: Moderate problems | 0 | 1
  Anxiety/depression: Severe problems | 0 | 1
  Anxiety/depression: Extreme problems | 0 | 0
  Anxiety/depression: Data missing | 1 | 4

26. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Intrathecal Drug Delivery Device (IDDD)-Related Adverse Events
Description: An adverse event (AE) was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product-related. Treatment-emergent AEs for the no IT treatment group were defined as all AEs occurring on or after the date of randomization and at or before the end of the study (EOS) visit. Treatment-emergent AEs for the IT treatment group were defined as all AEs occurring on or after the date of the first IDDD implant surgery or Treatment-Emergentfirst dose of the investigational product (whichever was earlier) and at or before the EOS visit (+30 days) or 2 weeks after the removal of the last IDDD (whichever was later).
Time Frame: From start of study treatment up to Week 53
Population: Safety population included all randomized participants with any post-randomization safety assessments, analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | No IT Treatment | IT Treatment
Number analyzed (Participants) | 15 | 33
Participants
  TEAEs | 14 | 33
  IDDD-related AE | 0 | 22

27. Secondary Outcome: Composite Scores of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The composite score for the cognitive scale, language scale, and motor scale are normed and have a mean=100, SD=15 and range of 40-160. Higher values denote stronger skills and abilities in the domain, indicating better outcomes. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: Score on a scale
Arm/Group | Substudy
Number analyzed (Participants) | 9
Score on a scale
  Baseline: Participant 1: Motor: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor | 97
  Week 16: Participant 1: Motor: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor | 82
  Week 28: Participant 1: Motor: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor | 67
  Week 40: Participant 1: Motor: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor | 94
  Week 52: Participant 1: Motor: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor | 79
  Baseline: Participant 2: Motor: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor | 82
  Week 16: Participant 2: Motor: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor | 76
  Week 28: Participant 2: Motor: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor | 82
  Week 40: Participant 2: Motor: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor | 76
  Baseline: Participant 3: Motor: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor | 82
  Week 16: Participant 3: Motor: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor | 79
  Week 28: Participant 3: Motor: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor | 88
  Week 40: Participant 3: Motor: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor | 88
  Week 52: Participant 3: Motor: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor | 82
  Baseline: Participant 4: Motor: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor | 76
  Week 16: Participant 4: Motor: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor | 91
  Week 28: Participant 4: Motor: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor | 91
  Baseline: Participant 5: Motor: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor | 94
  Week 16: Participant 5: Motor: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor | 67
  Week 28: Participant 5: Motor: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor | 85
  Baseline: Participant 6: Motor: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor | 103
  Week 16: Participant 6: Motor: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor | 107
  Week 28: Participant 6: Motor: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor | 103
  Week 40: Participant 6: Motor: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor | 107
  Week 52: Participant 6: Motor: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor | 85
  Baseline: Participant 7: Motor: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor | 85
  Week 16: Participant 7: Motor: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor | 76
  Week 28: Participant 7: Motor: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor | 79
  Week 40: Participant 7: Motor: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor | 79
  Baseline: Participant 8: Motor: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor | 91
  Week 16: Participant 8: Motor: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor | 91
  Week 28: Participant 8: Motor: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor | 88
  Baseline: Participant 9: Motor: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor | 85
  Week 16: Participant 9: Motor: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor | 88
  Week 28:Participant 9: Motor: number analyzed (Participants) | 1
  Week 28:Participant 9: Motor | 85
  Week 40: Participant 9: Motor: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor | 85
  Week 52: Participant 9: Motor: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor | 91
  Baseline: Participant 1: Language: number analyzed (Participants) | 1
  Baseline: Participant 1: Language | 91
  Week 16: Participant 1: Language: number analyzed (Participants) | 1
  Week 16: Participant 1: Language | 89
  Week 28: Participant 1: Language: number analyzed (Participants) | 1
  Week 28: Participant 1: Language | 91
  Week 40: Participant 1: Language: number analyzed (Participants) | 1
  Week 40: Participant 1: Language | 91
  Week 52: Participant 1: Language: number analyzed (Participants) | 1
  Week 52: Participant 1: Language | 94
  Baseline: Participant 2: Language: number analyzed (Participants) | 1
  Baseline: Participant 2: Language | 74
  Week 16: Participant 2: Language: number analyzed (Participants) | 1
  Week 16: Participant 2: Language | 77
  Week 28: Participant 2: Language: number analyzed (Participants) | 1
  Week 28: Participant 2: Language | 74
  Week 40: Participant 2: Language: number analyzed (Participants) | 1
  Week 40: Participant 2: Language | 79
  Baseline: Participant 3: Language: number analyzed (Participants) | 1
  Baseline: Participant 3: Language | 79
  Week 16: Participant 3: Language: number analyzed (Participants) | 1
  Week 16: Participant 3: Language | 77
  Week 28: Participant 3: Language: number analyzed (Participants) | 1
  Week 28: Participant 3: Language | 71
  Week 40: Participant 3: Language: number analyzed (Participants) | 1
  Week 40: Participant 3: Language | 91
  Week 52: Participant 3: Language: number analyzed (Participants) | 1
  Week 52: Participant 3: Language | 86
  Baseline: Participant 4: Language: number analyzed (Participants) | 1
  Baseline: Participant 4: Language | 79
  Week 16: Participant 4: Language: number analyzed (Participants) | 1
  Week 16: Participant 4: Language | 89
  Week 28: Participant 4: Language: number analyzed (Participants) | 1
  Week 28: Participant 4: Language | 89
  Baseline: Participant 5: Language: number analyzed (Participants) | 1
  Baseline: Participant 5: Language | 59
  Week 16: Participant 5: Language: number analyzed (Participants) | 1
  Week 16: Participant 5: Language | 53
  Week 28: Participant 5: Language: number analyzed (Participants) | 1
  Week 28: Participant 5: Language | 47
  Baseline: Participant 6: Language: number analyzed (Participants) | 1
  Baseline: Participant 6: Language | 89
  Week 16: Participant 6: Language: number analyzed (Participants) | 1
  Week 16: Participant 6: Language | 86
  Week 28: Participant 6: Language: number analyzed (Participants) | 1
  Week 28: Participant 6: Language | 77
  Week 40: Participant 6: Language: number analyzed (Participants) | 1
  Week 40: Participant 6: Language | 89
  Week 52: Participant 6: Language: number analyzed (Participants) | 1
  Week 52: Participant 6: Language | 83
  Baseline: Participant 7: Language: number analyzed (Participants) | 1
  Baseline: Participant 7: Language | 79
  Week 16: Participant 7: Language: number analyzed (Participants) | 1
  Week 16: Participant 7: Language | 74
  Week 28: Participant 7: Language: number analyzed (Participants) | 1
  Week 28: Participant 7: Language | 74
  Week 40: Participant 7: Language: number analyzed (Participants) | 1
  Week 40: Participant 7: Language | 71
  Baseline: Participant 8: Language: number analyzed (Participants) | 1
  Baseline: Participant 8: Language | 86
  Week 16: Participant 8: Language: number analyzed (Participants) | 1
  Week 16: Participant 8: Language | 100
  Week 28: Participant 8: Language: number analyzed (Participants) | 1
  Week 28: Participant 8: Language | 103
  Baseline: Participant 9: Language: number analyzed (Participants) | 1
  Baseline: Participant 9: Language | 62
  Week 16: Participant 9: Language: number analyzed (Participants) | 1
  Week 16: Participant 9: Language | 71
  Week 28: Participant 9: Language: number analyzed (Participants) | 1
  Week 28: Participant 9: Language | 71
  Week 40: Participant 9: Language: number analyzed (Participants) | 1
  Week 40: Participant 9: Language | 79
  Week 52: Participant 9: Language: number analyzed (Participants) | 1
  Week 52: Participant 9: Language | 74
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 85
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 90
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 90
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 100
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 95
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 75
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 90
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 90
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 85
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 90
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 85
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 90
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 90
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 85
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 80
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 95
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 100
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 85
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 85
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 80
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 80
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 100
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 95
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 105
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 90
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 85
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 90
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 85
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 80
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 90
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 100
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 110
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 85
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 90
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 90
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 90
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 95

28. Secondary Outcome: Percentile Scores of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. Percentile scores range from 1 to 99 with 50 as the mean and median. Higher percentile means higher the rank of the child relative to the normed population. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: Percentile score
Arm/Group | Substudy
Number analyzed (Participants) | 9
Percentile score
  Baseline: Participant 1: Motor: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor | 42
  Week 16: Participant 1: Motor: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor | 12
  Week 28: Participant 1: Motor: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor | 1
  Week 40: Participant 1: Motor: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor | 34
  Week 52: Participant 1: Motor: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor | 8
  Baseline: Participant 2: Motor: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor | 12
  Week 16: Participant 2: Motor: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor | 5
  Week 28: Participant 2: Motor: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor | 12
  Week 40: Participant 2: Motor: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor | 5
  Baseline: Participant 3: Motor: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor | 12
  Week 16: Participant 3: Motor: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor | 8
  Week 28: Participant 3: Motor: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor | 21
  Week 40: Participant 3: Motor: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor | 21
  Week 52: Participant 3: Motor: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor | 12
  Baseline: Participant 4: Motor: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor | 5
  Week 16: Participant 4: Motor: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor | 27
  Week 28: Participant 4: Motor: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor | 27
  Baseline: Participant 5: Motor: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor | 34
  Week 16: Participant 5: Motor: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor | 1
  Week 28: Participant 5: Motor: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor | 16
  Baseline: Participant 6: Motor: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor | 58
  Week 16: Participant 6: Motor: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor | 68
  Week 28: Participant 6: Motor: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor | 58
  Week 40: Participant 6: Motor: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor | 68
  Week 52: Participant 6: Motor: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor | 16
  Baseline: Participant 7: Motor: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor | 16
  Week 16: Participant 7: Motor: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor | 5
  Week 28: Participant 7: Motor: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor | 8
  Week 40: Participant 7: Motor: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor | 1
  Baseline: Participant 8: Motor: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor | 27
  Week 16: Participant 8: Motor: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor | 27
  Week 28: Participant 8: Motor: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor | 21
  Baseline: Participant 9: Motor: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor | 16
  Week 16: Participant 9: Motor: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor | 21
  Week 28: Participant 9: Motor: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor | 16
  Week 40: Participant 9: Motor: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor | 16
  Week 52: Participant 9: Motor: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor | 27
  Baseline: Participant 1: Language: number analyzed (Participants) | 1
  Baseline: Participant 1: Language | 27
  Week 16: Participant 1: Language: number analyzed (Participants) | 1
  Week 16: Participant 1: Language | 23
  Week 28: Participant 1: Language: number analyzed (Participants) | 1
  Week 28: Participant 1: Language | 27
  Week 40: Participant 1: Language: number analyzed (Participants) | 1
  Week 40: Participant 1: Language | 27
  Week 52: Participant 1: Language: number analyzed (Participants) | 1
  Week 52: Participant 1: Language | 34
  Baseline: Participant 2: Language: number analyzed (Participants) | 1
  Baseline: Participant 2: Language | 4
  Week 16: Participant 2: Language: number analyzed (Participants) | 1
  Week 16: Participant 2: Language | 6
  Week 28: Participant 2: Language: number analyzed (Participants) | 1
  Week 28: Participant 2: Language | 4
  Week 40: Participant 2: Language: number analyzed (Participants) | 1
  Week 40: Participant 2: Language | 8
  Baseline: Participant 3: Language: number analyzed (Participants) | 1
  Baseline: Participant 3: Language | 8
  Week 16: Participant 3: Language: number analyzed (Participants) | 1
  Week 16: Participant 3: Language | 6
  Week 28: Participant 3: Language: number analyzed (Participants) | 1
  Week 28: Participant 3: Language | 3
  Week 40: Participant 3: Language: number analyzed (Participants) | 1
  Week 40: Participant 3: Language | 27
  Week 52: Participant 3: Language: number analyzed (Participants) | 1
  Week 52: Participant 3: Language | 18
  Baseline: Participant 4: Language: number analyzed (Participants) | 1
  Baseline: Participant 4: Language | 8
  Week 16: Participant 4: Language: number analyzed (Participants) | 1
  Week 16: Participant 4: Language | 23
  Week 28: Participant 4: Language: number analyzed (Participants) | 1
  Week 28: Participant 4: Language | 23
  Baseline: Participant 5: Language: number analyzed (Participants) | 1
  Baseline: Participant 5: Language | 0.3
  Week 16: Participant 5: Language: number analyzed (Participants) | 1
  Week 16: Participant 5: Language | 0.1
  Week 28: Participant 5: Language: number analyzed (Participants) | 1
  Week 28: Participant 5: Language | 0.1
  Baseline: Participant 6: Language: number analyzed (Participants) | 1
  Baseline: Participant 6: Language | 23
  Week 16: Participant 6: Language: number analyzed (Participants) | 1
  Week 16: Participant 6: Language | 18
  Week 28: Participant 6: Language: number analyzed (Participants) | 1
  Week 28: Participant 6: Language | 6
  Week 40: Participant 6: Language: number analyzed (Participants) | 1
  Week 40: Participant 6: Language | 23
  Week 52: Participant 6: Language: number analyzed (Participants) | 1
  Week 52: Participant 6: Language | 13
  Baseline: Participant 7: Language: number analyzed (Participants) | 1
  Baseline: Participant 7: Language | 8
  Week 16: Participant 7: Language: number analyzed (Participants) | 1
  Week 16: Participant 7: Language | 4
  Week 28: Participant 7: Language: number analyzed (Participants) | 1
  Week 28: Participant 7: Language | 4
  Week 40: Participant 7: Language: number analyzed (Participants) | 1
  Week 40: Participant 7: Language | 3
  Baseline: Participant 8: Language: number analyzed (Participants) | 1
  Baseline: Participant 8: Language | 18
  Week 16: Participant 8: Language: number analyzed (Participants) | 1
  Week 16: Participant 8: Language | 50
  Week 28: Participant 8: Language: number analyzed (Participants) | 1
  Week 28: Participant 8: Language | 58
  Baseline: Participant 9: Language: number analyzed (Participants) | 1
  Baseline: Participant 9: Language | 1
  Week 16: Participant 9: Language: number analyzed (Participants) | 1
  Week 16: Participant 9: Language | 3
  Week 28: Participant 9: Language: number analyzed (Participants) | 1
  Week 28: Participant 9: Language | 3
  Week 40: Participant 9: Language: number analyzed (Participants) | 1
  Week 40: Participant 9: Language | 8
  Week 52: Participant 9: Language: number analyzed (Participants) | 1
  Week 52: Participant 9: Language | 4
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 16
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 25
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 25
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 50
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 37
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 5
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 25
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 25
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 16
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 25
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 16
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 25
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 25
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 16
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 9
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 37
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 50
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 16
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 16
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 9
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 9
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 50
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 37
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 63
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 25
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 16
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 25
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 16
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 9
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 25
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 50
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 75
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 16
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 25
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 25
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 25
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 37

29. Secondary Outcome: Age Equivalent Scores of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. Standardized scores (range 40-160) were converted to age- equivalent scores to measure ability, skill, and knowledge expressed as the age at which most individuals reach the same level (age norm; range: 0, unbound). Higher values present better outcomes. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: Score on a scale
Arm/Group | Substudy
Number analyzed (Participants) | 9
Score on a scale
  Baseline: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Fine | 28
  Baseline: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Gross | 24
  Week 16: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Fine | 28
  Week 16: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Gross | 20
  Week 28: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Fine | 18
  Week 28: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Gross | 21
  Week 40: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Fine | 32
  Week 40: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Gross | 38
  Week 52: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Fine | 34
  Week 52: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Gross | 24
  Baseline: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Fine | 25
  Baseline: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Gross | 20
  Week 16: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Fine | 28
  Week 16: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Gross | 18
  Week 28: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Fine | 32
  Week 28: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Gross | 24
  Week 40: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Fine | 29
  Week 40: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Gross | 23
  Baseline: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Fine | 26
  Baseline: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Gross | 18
  Week 16: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Fine | 26
  Week 16: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Gross | 21
  Week 28: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Fine | 32
  Week 28: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Gross | 31
  Week 40: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Fine | 32
  Week 40: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Gross | 29
  Week 52: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Fine | 29
  Week 52: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Gross | 29
  Baseline: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Fine | 29
  Baseline: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Gross | 19
  Week 16: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Fine | 33
  Week 16: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Gross | 38
  Week 28: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Fine | 31
  Week 28: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Gross | 41
  Baseline: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Fine | 28
  Baseline: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Gross | 27
  Week 16: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Fine | 25
  Week 16: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Gross | 20
  Week 28: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Fine | 29
  Week 28: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Gross | 31
  Week 40: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Fine | 26
  Week 40: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Gross | 27
  Week 52: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Fine | 28
  Week 52: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Gross | 35
  Baseline: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Fine | 16
  Baseline: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Gross | 15
  Week 16: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Fine | 25
  Week 16: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Gross | 20
  Week 28: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Fine | 26
  Week 28: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Gross | 23
  Week 40: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Fine | 31
  Week 40: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Gross | 26
  Week 52: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Fine | 25
  Week 52: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Gross | 20
  Baseline: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Fine | 26
  Baseline: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Gross | 20
  Week 16: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Fine | 25
  Week 16: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Gross | 23
  Week 28: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Fine | 28
  Week 28: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Gross | 24
  Week 40: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Fine | 29
  Week 40: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Gross | 27
  Week 52: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Fine | 29
  Week 52: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Gross | 31
  Baseline: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Fine | 31
  Baseline: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Gross | 31
  Week 16: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Fine | 38
  Week 16: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Gross | 31
  Week 28: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Fine | 35
  Week 28: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Gross | 31
  Baseline: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Fine | 25
  Baseline: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Gross | 18
  Week 16: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Fine | 27
  Week 16: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Gross | 21
  Week 28: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Fine | 31
  Week 28: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Gross | 20
  Week 40: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Fine | 31
  Week 40: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Gross | 26
  Week 52: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Fine | 34
  Week 52: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Gross | 31
  Baseline: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Receptive | 22
  Baseline: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Expressive | 25
  Week 16: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Receptive | 24
  Week 16: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Expressive | 27
  Week 28: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Receptive | 26
  Week 28: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Expressive | 33
  Week 40: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Receptive | 30
  Week 40: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Expressive | 33
  Week 52: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Receptive | 32
  Week 52: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Expressive | 34
  Baseline: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Receptive | 19
  Baseline: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Expressive | 18
  Week 16: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Receptive | 23
  Week 16: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Expressive | 19
  Week 28: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Receptive | 20
  Week 28: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Expressive | 24
  Week 40: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Receptive | 26
  Week 40: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Expressive | 25
  Baseline: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Receptive | 19
  Baseline: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Expressive | 19
  Week 16: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Receptive | 19
  Week 16: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Expressive | 23
  Week 28: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Receptive | 21
  Week 28: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Expressive | 22
  Week 40: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Receptive | 29
  Week 40: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Expressive | 33
  Week 52: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Receptive | 29
  Week 52: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Expressive | 29
  Baseline: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Receptive | 21
  Baseline: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Expressive | 25
  Week 16: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Receptive | 32
  Week 16: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Expressive | 30
  Week 28: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Receptive | 28
  Week 28: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Expressive | 38
  Baseline: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Receptive | 11
  Baseline: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Expressive | 12
  Week 16: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Receptive | 11
  Week 16: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Expressive | 7
  Week 28: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Receptive | 0.52
  Week 28: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Expressive | 7
  Week 40: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Receptive | 11
  Week 40: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Expressive | 13
  Week 52: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Receptive | 11
  Week 52: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Expressive | 10
  Baseline: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Receptive | 14
  Baseline: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Expressive | 12
  Week 16: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Receptive | 19
  Week 16: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Expressive | 16
  Week 28: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Receptive | 19
  Week 28: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Expressive | 14
  Week 40: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Receptive | 25
  Week 40: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Expressive | 19
  Week 52: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Receptive | 24
  Week 52: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Expressive | 19
  Baseline: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Receptive | 19
  Baseline: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Expressive | 21
  Week 16: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Receptive | 16
  Week 16: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Expressive | 23
  Week 28: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Receptive | 18
  Week 28: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Expressive | 25
  Week 40: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Receptive | 18
  Week 40: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Expressive | 24
  Week 52: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Receptive | 19
  Week 52: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Expressive | 22
  Baseline: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Receptive | 29
  Baseline: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Expressive | 26
  Week 16: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Receptive | 42
  Week 16: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Expressive | 38
  Week 28: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Receptive | 42
  Week 28: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Expressive | 34
  Baseline: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Receptive | 18
  Baseline: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Expressive | 5
  Week 16: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Receptive | 25
  Week 16: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Expressive | 2
  Week 28: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Receptive | 28
  Week 28: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Expressive | 7
  Week 40: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Receptive | 35
  Week 40: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Expressive | 16
  Week 52: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Receptive | 30
  Week 52: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Expressive | 17
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 22
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 26
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 30
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 38
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 36
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 21
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 28
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 29
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 28
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 24
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 25
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 28
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 28
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 29
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 23
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 36
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 41
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 23
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 27
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 25
  Week 40: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 5: Cognitive | 28
  Week 52: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 5: Cognitive | 28
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 12
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 21
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 22
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 28
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 25
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 24
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 27
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 27
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 27
  Week 52: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 7: Cognitive | 27
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 29
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 41
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 42
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 22
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 25
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 27
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 27
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 33

30. Secondary Outcome: Chronological Age of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. Chronological age of the participants when assessed by the BSID-III scale was reported. Range 16.59 - 45.21 months. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: Months
Arm/Group | Substudy
Number analyzed (Participants) | 9
Months
  Baseline: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Fine | 29.31
  Baseline: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Gross | 29.31
  Week 16: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Fine | 32.92
  Week 16: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Gross | 32.92
  Week 28: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Fine | 35.91
  Week 28: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Gross | 35.91
  Week 40: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Fine | 38.90
  Week 40: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Gross | 38.90
  Week 52: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Fine | 41.49
  Week 52: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Gross | 41.49
  Baseline: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Fine | 30.32
  Baseline: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Gross | 30.32
  Week 16: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Fine | 34.00
  Week 16: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Gross | 34.00
  Week 28: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Fine | 37.16
  Week 28: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Gross | 37.16
  Week 40: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Fine | 40.21
  Week 40: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Gross | 40.21
  Baseline: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Fine | 28.29
  Baseline: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Gross | 28.29
  Week 16: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Fine | 33.97
  Week 16: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Gross | 33.97
  Week 28: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Fine | 36.99
  Week 28: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Gross | 36.99
  Week 40: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Fine | 39.33
  Week 40: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Gross | 39.33
  Week 52: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Fine | 42.32
  Week 52: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Gross | 42.32
  Baseline: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Fine | 35.68
  Baseline: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Gross | 35.68
  Week 16: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Fine | 39.82
  Week 16: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Gross | 39.82
  Week 28: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Fine | 42.32
  Week 28: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Gross | 42.32
  Baseline: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Fine | 31.44
  Baseline: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Gross | 31.44
  Week 16: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Fine | 37.09
  Week 16: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Gross | 37.09
  Week 28: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Fine | 39.92
  Week 28: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Gross | 39.92
  Week 40: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Fine | 42.64
  Week 40: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Gross | 42.64
  Week 52: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Fine | 45.21
  Week 52: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Gross | 45.21
  Baseline: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Fine | 16.59
  Baseline: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Gross | 16.59
  Week 16: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Fine | 21.09
  Week 16: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Gross | 21.09
  Week 28: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Fine | 23.72
  Week 28: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Gross | 23.72
  Week 40: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Fine | 26.61
  Week 40: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Gross | 26.61
  Week 52: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Fine | 29.14
  Week 52: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Gross | 29.14
  Baseline: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Fine | 30.09
  Baseline: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Gross | 30.09
  Week 16: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Fine | 35.12
  Week 16: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Gross | 35.12
  Week 28: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Fine | 37.88
  Week 28: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Gross | 37.88
  Week 40: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Fine | 40.87
  Week 40: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Gross | 40.87
  Week 52: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Fine | 43.56
  Week 52: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Gross | 43.56
  Baseline: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Fine | 35.61
  Baseline: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Gross | 35.61
  Week 16: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Fine | 39.82
  Week 16: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Gross | 39.82
  Week 28: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Fine | 42.35
  Week 28: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Gross | 42.35
  Baseline: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Fine | 26.25
  Baseline: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Gross | 26.25
  Week 16: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Fine | 30.03
  Week 16: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Gross | 30.03
  Week 28: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Fine | 33.25
  Week 28: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Gross | 33.25
  Week 40: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Fine | 36.11
  Week 40: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Gross | 36.11
  Week 52: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Fine | 38.64
  Week 52: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Gross | 38.64
  Baseline: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Receptive | 29.31
  Baseline: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Expressive | 29.31
  Week 16: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Receptive | 32.92
  Week 16: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Expressive | 32.92
  Week 28: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Receptive | 35.91
  Week 28: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Expressive | 35.91
  Week 40: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Receptive | 38.90
  Week 40: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Expressive | 38.90
  Week 52: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Receptive | 41.49
  Week 52: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Expressive | 41.49
  Baseline: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Receptive | 30.32
  Baseline: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Expressive | 30.32
  Week 16: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Receptive | 34.00
  Week 16: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Expressive | 34.00
  Week 28: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Receptive | 37.16
  Week 28: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Expressive | 37.16
  Week 40: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Receptive | 40.21
  Week 40: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Expressive | 40.21
  Baseline: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Receptive | 28.29
  Baseline: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Expressive | 28.29
  Week 16: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Receptive | 33.97
  Week 16: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Expressive | 33.97
  Week 28: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Receptive | 36.99
  Week 28: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Expressive | 36.99
  Week 40: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Receptive | 39.33
  Week 40: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Expressive | 39.33
  Week 52: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Receptive | 42.32
  Week 52: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Expressive | 42.32
  Baseline: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Receptive | 35.68
  Baseline: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Expressive | 35.68
  Week 16: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Receptive | 39.82
  Week 16: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Expressive | 39.82
  Week 28: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Receptive | 42.32
  Week 28: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Expressive | 42.32
  Baseline: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Receptive | 31.44
  Baseline: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Expressive | 31.44
  Week 16: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Receptive | 37.09
  Week 16: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Expressive | 37.09
  Week 28: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Receptive | 39.92
  Week 28: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Expressive | 39.92
  Week 40: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Receptive | 42.64
  Week 40: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Expressive | 42.64
  Week 52: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Receptive | 45.21
  Week 52: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Expressive | 45.21
  Baseline: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Receptive | 16.59
  Baseline: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Expressive | 16.59
  Week 16: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Receptive | 21.09
  Week 16: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Expressive | 21.09
  Week 28: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Receptive | 23.72
  Week 28: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Expressive | 23.72
  Week 40: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Receptive | 26.61
  Week 40: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Expressive | 26.61
  Week 52: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Receptive | 29.14
  Week 52: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Expressive | 29.14
  Baseline: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Receptive | 30.09
  Baseline: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Expressive | 30.09
  Week 16: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Receptive | 35.12
  Week 16: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Expressive | 35.12
  Week 28: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Receptive | 37.88
  Week 28: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Expressive | 37.88
  Week 40: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Receptive | 40.87
  Week 40: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Expressive | 40.87
  Week 52: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Receptive | 43.56
  Week 52: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Expressive | 43.56
  Baseline: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Receptive | 35.61
  Baseline: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Expressive | 35.61
  Week 16: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Receptive | 39.82
  Week 16: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Expressive | 39.82
  Week 28: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Receptive | 42.35
  Week 28: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Expressive | 42.35
  Baseline: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Receptive | 26.25
  Baseline: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Expressive | 26.25
  Week 16: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Receptive | 30.03
  Week 16: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Expressive | 30.03
  Week 28: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Receptive | 33.25
  Week 28: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Expressive | 33.25
  Week 40: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Receptive | 36.11
  Week 40: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Expressive | 36.11
  Week 52: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Receptive | 38.64
  Week 52: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Expressive | 38.64
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 29.31
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 32.92
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 35.91
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 38.90
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 41.49
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 30.32
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 34.00
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 37.16
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 40.21
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 28.29
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 33.97
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 36.99
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 39.33
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 42.32
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 35.68
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 39.82
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 42.32
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 31.44
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 37.09
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 39.92
  Week 40: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 5: Cognitive | 42.64
  Week 52: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 5: Cognitive | 45.21
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 16.59
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 21.09
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 23.72
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 26.61
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 29.14
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 30.09
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 35.12
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 37.88
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 40.87
  Week 52: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 7: Cognitive | 43.56
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 35.61
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 39.82
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 42.35
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 26.25
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 30.03
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 33.25
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 36.11
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 38.64

31. Secondary Outcome: Development Quotient (DQ) of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. The development quotient (DQ) is a means to express a neurodevelopmental/cognitive delay which will be computed as a ratio and expressed as a percentage using the age equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0-100). Higher values present better outcomes. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: Percentage of chronological age
Arm/Group | Substudy
Number analyzed (Participants) | 9
Percentage of chronological age
  Baseline: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Fine | 95.5
  Baseline: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Gross | 81.9
  Week 16: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Fine | 85.1
  Week 16: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Gross | 60.8
  Week 28: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Fine | 50.1
  Week 28: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Gross | 58.5
  Week 40: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Fine | 82.3
  Week 40: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Gross | 97.7
  Week 52: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Fine | 81.9
  Week 52: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Gross | 57.8
  Baseline: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Fine | 82.4
  Baseline: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Gross | 66
  Week 16: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Fine | 82.3
  Week 16: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Gross | 52.9
  Week 28: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Fine | 86.1
  Week 28: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Gross | 64.6
  Week 40: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Fine | 72.1
  Week 40: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Gross | 57.2
  Baseline: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Fine | 91.9
  Baseline: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Gross | 63.6
  Week 16: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Fine | 76.5
  Week 16: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Gross | 61.8
  Week 28: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Fine | 86.5
  Week 28: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Gross | 83.8
  Week 40: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Fine | 81.4
  Week 40: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Gross | 73.7
  Week 52: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Fine | 68.5
  Week 52: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Gross | 68.5
  Baseline: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Fine | 81.3
  Baseline: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Gross | 53.3
  Week 16: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Fine | 82.9
  Week 16: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Gross | 95.4
  Week 28: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Fine | 73.3
  Week 28: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Gross | 96.9
  Baseline: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Fine | 89.1
  Baseline: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Gross | 85.9
  Week 16: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Fine | 67.4
  Week 16: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Gross | 53.9
  Week 28: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Fine | 72.6
  Week 28: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Gross | 77.7
  Week 40: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Fine | 61
  Week 40: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Gross | 63.3
  Week 52: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Fine | 61.9
  Week 52: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Gross | 77.4
  Baseline: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Fine | 96.4
  Baseline: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Gross | 90.4
  Week 16: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Fine | 118.5
  Week 16: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Gross | 94.8
  Week 28: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Fine | 109.6
  Week 28: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Gross | 97
  Week 40: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Fine | 116.5
  Week 40: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Gross | 97.7
  Week 52: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Fine | 85.8
  Week 52: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Gross | 68.6
  Baseline: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Fine | 86.4
  Baseline: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Gross | 66.5
  Week 16: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Fine | 71.2
  Week 16: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Gross | 65.5
  Week 28: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Fine | 73.9
  Week 28: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Gross | 63.4
  Week 40: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Fine | 71
  Week 40: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Gross | 66.1
  Week 52: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Fine | 66.6
  Week 52: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Gross | 71.2
  Baseline: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Fine | 87
  Baseline: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Gross | 87
  Week 16: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Fine | 95.4
  Week 16: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Gross | 77.9
  Week 28: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Fine | 82.6
  Week 28: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Gross | 73.2
  Baseline: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Fine | 95.2
  Baseline: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Gross | 68.6
  Week 16: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Fine | 89.9
  Week 16: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Gross | 69.9
  Week 28: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Fine | 93.2
  Week 28: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Gross | 60.2
  Week 40: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Fine | 85.9
  Week 40: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Gross | 72
  Week 52: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Fine | 88
  Week 52: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Gross | 80.2
  Baseline: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Receptive | 75.1
  Baseline: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Expressive | 85.3
  Week 16: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Receptive | 72.9
  Week 16: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Expressive | 82
  Week 28: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Receptive | 72.4
  Week 28: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Expressive | 91.9
  Week 40: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Receptive | 77.1
  Week 40: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Expressive | 84.8
  Week 52: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Receptive | 77.1
  Week 52: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Expressive | 81.9
  Baseline: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Receptive | 62.7
  Baseline: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Expressive | 59.4
  Week 16: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Receptive | 67.6
  Week 16: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Expressive | 55.9
  Week 28: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Receptive | 53.8
  Week 28: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Expressive | 64.6
  Week 40: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Receptive | 64.7
  Week 40: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Expressive | 62.2
  Baseline: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Receptive | 67.2
  Baseline: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Expressive | 67.2
  Week 16: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Receptive | 55.9
  Week 16: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Expressive | 67.7
  Week 28: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Receptive | 56.8
  Week 28: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Expressive | 59.5
  Week 40: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Receptive | 73.7
  Week 40: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Expressive | 83.9
  Week 52: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Receptive | 68.5
  Week 52: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Expressive | 68.5
  Baseline: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Receptive | 58.9
  Baseline: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Expressive | 70.1
  Week 16: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Receptive | 80.4
  Week 16: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Expressive | 75.3
  Week 28: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Receptive | 66.2
  Week 28: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Expressive | 89.8
  Baseline: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Receptive | 35
  Baseline: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Expressive | 38.2
  Week 16: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Receptive | 29.7
  Week 16: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Expressive | 18.9
  Week 28: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Receptive | 1.3
  Week 28: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Expressive | 17.5
  Week 40: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Receptive | 25.8
  Week 40: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Expressive | 30.5
  Week 52: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Receptive | 24.3
  Week 52: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Expressive | 22.1
  Baseline: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Receptive | 84.4
  Baseline: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Expressive | 72.3
  Week 16: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Receptive | 90.1
  Week 16: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Expressive | 75.9
  Week 28: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Receptive | 80.1
  Week 28: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Expressive | 59
  Week 40: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Receptive | 93.9
  Week 40: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Expressive | 71.4
  Week 52: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Receptive | 82.4
  Week 52: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Expressive | 65.2
  Baseline: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Receptive | 63.1
  Baseline: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Expressive | 69.8
  Week 16: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Receptive | 45.6
  Week 16: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Expressive | 65.5
  Week 28: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Receptive | 47.5
  Week 28: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Expressive | 66
  Week 40: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Receptive | 44
  Week 40: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Expressive | 58.7
  Week 52: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Receptive | 43.6
  Week 52: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Expressive | 50.5
  Baseline: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Receptive | 81.4
  Baseline: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Expressive | 73
  Week 16: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Receptive | 105.5
  Week 16: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Expressive | 95.4
  Week 28: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Receptive | 99.2
  Week 28: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Expressive | 80.3
  Baseline: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Receptive | 68.6
  Baseline: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Expressive | 19
  Week 16: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Receptive | 83.3
  Week 16: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Expressive | 6.7
  Week 28: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Receptive | 84.2
  Week 28: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Expressive | 21.1
  Week 40: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Receptive | 96.9
  Week 40: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Expressive | 44.3
  Week 52: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Receptive | 77.6
  Week 52: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Expressive | 44
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 75.1
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 79
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 83.5
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 97.7
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 86.8
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 69.3
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 82.3
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 78
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 69.6
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 84.8
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 73.6
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 75.7
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 71.2
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 68.5
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 64.5
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 90.4
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 96.9
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 73.2
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 72.8
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 62.6
  Week 40: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 5: Cognitive | 65.7
  Week 52: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 5: Cognitive | 61.9
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 72.3
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 99.6
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 92.7
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 105.2
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 85.8
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 79.7
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 76.9
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 71.3
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 66.1
  Week 52: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 7: Cognitive | 62
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 81.4
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 103
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 99.2
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 83.8
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 83.3
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 81.2
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 74.8
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 85.4

32. Secondary Outcome: Raw Scores of Bayley Scales of Infant Development (BSID-III) Scale in Substudy Population
Description: Participants who were younger than 3 years were assessed using the BSID-III. The BSID--III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. Raw scores are converted to scaled scores that are based on normed populations. Raw score ranges: Cognitive scale 0-91, Receptive communication 0-49, Expressive communication 0-48, Fine motor 0-66 and Gross motor 0-72. Higher values indicate better outcomes. Participant wise data at evaluable timepoints was reported for this outcome.
Time Frame: Baseline up to Week 52
Population: Substudy population included all participants enrolled and treated with investigational product in the substudy.
Measure: Number; unit: score on a scale
Arm/Group | Substudy
Number analyzed (Participants) | 9
score on a scale
  Baseline: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Fine | 42
  Baseline: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 1: Motor-Gross | 57
  Week 16: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Fine | 42
  Week 16: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 1: Motor-Gross | 54
  Week 28: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Fine | 34
  Week 28: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 1: Motor-Gross | 55
  Week 40: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Fine | 45
  Week 40: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 1: Motor-Gross | 65
  Week 52: Participant 1: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Fine | 47
  Week 52: Participant 1: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 1: Motor-Gross | 57
  Baseline: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Fine | 39
  Baseline: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 2: Motor-Gross | 54
  Week 16: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Fine | 42
  Week 16: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 2: Motor-Gross | 52
  Week 28: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Fine | 45
  Week 28: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 2: Motor-Gross | 57
  Week 40: Participant 2: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Fine | 43
  Week 40: Participant 2: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 2: Motor-Gross | 56
  Baseline: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Fine | 40
  Baseline: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 3: Motor-Gross | 51
  Week 16: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Fine | 40
  Week 16: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 3: Motor-Gross | 55
  Week 28: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Fine | 45
  Week 28: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 3: Motor-Gross | 61
  Week 40: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Fine | 45
  Week 40: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 3: Motor-Gross | 60
  Week 52: Participant 3: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Fine | 43
  Week 52: Participant 3: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 3: Motor-Gross | 60
  Baseline: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Fine | 43
  Baseline: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 4: Motor-Gross | 53
  Week 16: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Fine | 46
  Week 16: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 4: Motor-Gross | 64
  Week 28: Participant 4: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Fine | 44
  Week 28: Participant 4: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 4: Motor-Gross | 66
  Baseline: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Fine | 42
  Baseline: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 5: Motor-Gross | 59
  Week 16: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Fine | 39
  Week 16: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 5: Motor-Gross | 54
  Week 28: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Fine | 43
  Week 28: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 5: Motor-Gross | 61
  Week 40: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Fine | 40
  Week 40: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 5: Motor-Gross | 59
  Week 52: Participant 5: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Fine | 42
  Week 52: Participant 5: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 5: Motor-Gross | 63
  Baseline: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Fine | 32
  Baseline: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 6: Motor-Gross | 47
  Week 16: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Fine | 39
  Week 16: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 6: Motor-Gross | 54
  Week 28: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Fine | 40
  Week 28: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 6: Motor-Gross | 56
  Week 40: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Fine | 44
  Week 40: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 6: Motor-Gross | 58
  Week 52: Participant 6: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Fine | 39
  Week 52: Participant 6: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 6: Motor-Gross | 54
  Baseline: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Fine | 40
  Baseline: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 7: Motor-Gross | 54
  Week 16: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Fine | 39
  Week 16: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 7: Motor-Gross | 56
  Week 28: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Fine | 42
  Week 28: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 7: Motor-Gross | 57
  Week 40: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Fine | 43
  Week 40: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 7: Motor-Gross | 59
  Week 52: Participant 7: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Fine | 43
  Week 52: Participant 7: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 7: Motor-Gross | 61
  Baseline: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Fine | 44
  Baseline: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 8: Motor-Gross | 61
  Week 16: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Fine | 50
  Week 16: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 8: Motor-Gross | 61
  Week 28: Participant 8: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Fine | 48
  Week 28: Participant 8: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 8: Motor-Gross | 61
  Baseline: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Fine | 39
  Baseline: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Baseline: Participant 9: Motor-Gross | 51
  Week 16: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Fine | 41
  Week 16: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 16: Participant 9: Motor-Gross | 55
  Week 28: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Fine | 44
  Week 28: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 28: Participant 9: Motor-Gross | 54
  Week 40: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Fine | 44
  Week 40: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 40: Participant 9: Motor-Gross | 58
  Week 52: Participant 9: Motor-Fine: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Fine | 47
  Week 52: Participant 9: Motor-Gross: number analyzed (Participants) | 1
  Week 52: Participant 9: Motor-Gross | 61
  Baseline: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Receptive | 25
  Baseline: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 1: Language-Expressive | 31
  Week 16: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Receptive | 27
  Week 16: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 1: Language-Expressive | 33
  Week 28: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Receptive | 29
  Week 28: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 1: Language-Expressive | 37
  Week 40: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Receptive | 32
  Week 40: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 1: Language-Expressive | 37
  Week 52: Participant 1: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Receptive | 34
  Week 52: Participant 1: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 1: Language-Expressive | 38
  Baseline: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Receptive | 21
  Baseline: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 2: Language-Expressive | 22
  Week 16: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Receptive | 26
  Week 16: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 2: Language-Expressive | 24
  Week 28: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Receptive | 23
  Week 28: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 2: Language-Expressive | 30
  Week 40: Participant 2: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Receptive | 29
  Week 40: Participant 2: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 2: Language-Expressive | 31
  Baseline: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Receptive | 22
  Baseline: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 3: Language-Expressive | 24
  Week 16: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Receptive | 21
  Week 16: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 3: Language-Expressive | 29
  Week 28: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Receptive | 24
  Week 28: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 3: Language-Expressive | 28
  Week 40: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Receptive | 31
  Week 40: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 3: Language-Expressive | 37
  Week 52: Participant 3: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Receptive | 31
  Week 52: Participant 3: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 3: Language-Expressive | 34
  Baseline: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Receptive | 24
  Baseline: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 4: Language-Expressive | 31
  Week 16: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Receptive | 34
  Week 16: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 4: Language-Expressive | 35
  Week 28: Participant 4: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Receptive | 30
  Week 28: Participant 4: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 4: Language-Expressive | 40
  Baseline: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Receptive | 14
  Baseline: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 5: Language-Expressive | 14
  Week 16: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Receptive | 14
  Week 16: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 5: Language-Expressive | 9
  Week 28: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Receptive | 2
  Week 28: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 5: Language-Expressive | 9
  Week 40: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Receptive | 14
  Week 40: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 5: Language-Expressive | 16
  Week 52: Participant 5: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Receptive | 14
  Week 52: Participant 5: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 5: Language-Expressive | 12
  Baseline: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Receptive | 16
  Baseline: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 6: Language-Expressive | 14
  Week 16: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Receptive | 21
  Week 16: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 6: Language-Expressive | 19
  Week 28: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Receptive | 21
  Week 28: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 6: Language-Expressive | 17
  Week 40: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Receptive | 28
  Week 40: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 6: Language-Expressive | 23
  Week 52: Participant 6: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Receptive | 27
  Week 52: Participant 6: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 6: Language-Expressive | 24
  Baseline: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Receptive | 21
  Baseline: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 7: Language-Expressive | 27
  Week 16: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Receptive | 18
  Week 16: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 7: Language-Expressive | 29
  Week 28: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Receptive | 20
  Week 28: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 7: Language-Expressive | 31
  Week 40: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Receptive | 20
  Week 40: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 7: Language-Expressive | 30
  Week 52: Participant 7: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Receptive | 21
  Week 52: Participant 7: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 7: Language-Expressive | 28
  Baseline: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Receptive | 31
  Baseline: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 8: Language-Expressive | 32
  Week 16: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Receptive | 40
  Week 16: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 8: Language-Expressive | 40
  Week 28: Participant 8: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Receptive | 42
  Week 28: Participant 8: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 8: Language-Expressive | 38
  Baseline: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Receptive | 20
  Baseline: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Baseline: Participant 9: Language-Expressive | 7
  Week 16: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Receptive | 28
  Week 16: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 16: Participant 9: Language-Expressive | 5
  Week 28: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Receptive | 30
  Week 28: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 28: Participant 9: Language-Expressive | 9
  Week 40: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Receptive | 36
  Week 40: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 40: Participant 9: Language-Expressive | 19
  Week 52: Participant 9: Language-Receptive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Receptive | 32
  Week 52: Participant 9: Language-Expressive: number analyzed (Participants) | 1
  Week 52: Participant 9: Language-Expressive | 21
  Baseline: Participant 1: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 1: Cognitive | 60
  Week 16: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 1: Cognitive | 66
  Week 28: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 1: Cognitive | 71
  Week 40: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 1: Cognitive | 78
  Week 52: Participant 1: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 1: Cognitive | 77
  Baseline: Participant 2: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 2: Cognitive | 57
  Week 16: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 2: Cognitive | 69
  Week 28: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 2: Cognitive | 70
  Week 40: Participant 2: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 2: Cognitive | 69
  Baseline: Participant 3: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 3: Cognitive | 63
  Week 16: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 3: Cognitive | 64
  Week 28: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 3: Cognitive | 69
  Week 40: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 3: Cognitive | 69
  Week 52: Participant 3: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 3: Cognitive | 70
  Baseline: Participant 4: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 4: Cognitive | 62
  Week 16: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 4: Cognitive | 77
  Week 28: Participant 4: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 4: Cognitive | 79
  Baseline: Participant 5: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 5: Cognitive | 62
  Week 16: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 5: Cognitive | 67
  Week 28: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 5: Cognitive | 65
  Week 40: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 5: Cognitive | 69
  Week 52: Participant 5: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 5: Cognitive | 69
  Baseline: Participant 6: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 6: Cognitive | 40
  Week 16: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 6: Cognitive | 58
  Week 28: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 6: Cognitive | 60
  Week 40: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 6: Cognitive | 69
  Week 52: Participant 6: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 6: Cognitive | 64
  Baseline: Participant 7: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 7: Cognitive | 63
  Week 16: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 7: Cognitive | 68
  Week 28: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 7: Cognitive | 68
  Week 40: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 7: Cognitive | 67
  Week 52: Participant 7: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 7: Cognitive | 67
  Baseline: Participant 8: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 8: Cognitive | 70
  Week 16: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 8: Cognitive | 79
  Week 28: Participant 8: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 8: Cognitive | 82
  Baseline: Participant 9: Cognitive: number analyzed (Participants) | 1
  Baseline: Participant 9: Cognitive | 59
  Week 16: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 16: Participant 9: Cognitive | 65
  Week 28: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 28: Participant 9: Cognitive | 67
  Week 40: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 40: Participant 9: Cognitive | 68
  Week 52: Participant 9: Cognitive: number analyzed (Participants) | 1
  Week 52: Participant 9: Cognitive | 74

ADVERSE EVENTS:
Time Frame: From start of study treatment up to Week 53
Description: For IT Treatment group 34 participants were randomized but only 33 participants are part of the safety population as 1 participant discontinued the study without receiving study treatment.
Arm/Group | No IT Treatment | IT Treatment | Substudy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/33 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/15 | 12/33 | 7/9
Other Adverse Events (participants affected / at risk) | 14/15 | 33/33 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No IT Treatment (N=15) | IT Treatment (N=33) | Substudy (N=9)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1) | 1 (1)
Device failure (General disorders) | 0 (0) | 2 (2) | 0 (0)
Device kink (General disorders) | 0 (0) | 3 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site effusion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 1 (2)
Vascular complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CSF cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 4 (5) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No IT Treatment (N=15) | IT Treatment (N=33) | Substudy (N=9)
Hypochromasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Toe walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 1 (1) | 4 (7) | 0 (0)
Diastolic hypotension (Vascular disorders) | 1 (1) | 4 (6) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Systolic hypertension (Vascular disorders) | 1 (1) | 4 (9) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 2 (11) | 2 (2) | 2 (7)
Astigmatism (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Excessive eye blinking (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 4 (4) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 10 (20) | 7 (8)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 25 (72) | 8 (27)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 2 (3) | 1 (1)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 2 (3)
Device breakage (General disorders) | 0 (0) | 2 (2) | 0 (0)
Device component issue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 0 (0) | 1 (1) | 1 (1)
Device kink (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 1 (2) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 4 (4) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Implant site effusion (General disorders) | 0 (0) | 6 (8) | 2 (3)
Implant site pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Implant site swelling (General disorders) | 0 (0) | 3 (3) | 0 (0)
Irritability (General disorders) | 0 (0) | 4 (4) | 2 (2)
Medical device complication (General disorders) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (3) | 3 (3)
Puncture site pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (10) | 19 (39) | 8 (17)
Vascular complication associated with device (General disorders) | 3 (8) | 5 (5) | 2 (7)
Congenital osteodystrophy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 4 (10) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (4) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 4 (7) | 9 (10) | 3 (8)
Ear infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 5 (6) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hand-Foot-And-Mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 13 (22) | 2 (4)
Otitis media (Infections and infestations) | 1 (1) | 4 (4) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (3)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 11 (15) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 2 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 14 (15) | 6 (8)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 4 (6) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 0 (0)
Albumin CSF increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 3 (3) | 8 (26) | 4 (20)
Blood pressure diastolic increased (Investigations) | 2 (2) | 6 (10) | 3 (3)
Blood pressure increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1) | 7 (20) | 4 (18)
Blood pressure systolic increased (Investigations) | 2 (3) | 7 (20) | 4 (15)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (2) | 2 (2) | 1 (1)
Body temperature decreased (Investigations) | 0 (0) | 5 (6) | 4 (5)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CSF cell count increased (Investigations) | 0 (0) | 4 (5) | 3 (5)
CSF glucose decreased (Investigations) | 1 (1) | 7 (9) | 2 (3)
CSF mononuclear cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CSF pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
CSF protein increased (Investigations) | 2 (2) | 5 (6) | 2 (2)
CSF white blood cell count increased (Investigations) | 0 (0) | 2 (2) | 1 (2)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 3 (4) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 5 (7) | 4 (4)
Eosinophil percentage increased (Investigations) | 0 (0) | 2 (3) | 2 (2)
Gamma-Glutamyltransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 2 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Heart rate decreased (Investigations) | 3 (5) | 7 (25) | 4 (17)
Heart rate increased (Investigations) | 4 (6) | 7 (17) | 4 (9)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 2 (2) | 4 (5) | 4 (13)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 1 (1)
Red blood cells CSF positive (Investigations) | 0 (0) | 3 (3) | 0 (0)
Respiratory rate decreased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
X-Ray abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (5)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 12 (23) | 3 (5)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1) | 5 (5) | 0 (0)
Subdural effusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (2) | 4 (4) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Communication disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphemia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Social avoidant behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 15 (33) | 4 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (10) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (10) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (5) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonmentor termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (7):
  • Study Protocol: original (2013-04-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_000.pdf
  • Study Protocol: Amendment 1 (2013-08-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_001.pdf
  • Study Protocol: Amendment 2 (2013-12-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_002.pdf
  • Study Protocol: Amendment 3 (2015-02-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_003.pdf
  • Study Protocol: Amendment 4 (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_004.pdf
  • Study Protocol: Amendment 5 (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/Prot_005.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02055118/SAP_006.pdf